| DIVISION | : Worldwide Development |
|---|---|
| Information Type : Reporting and Analysis Plan (RAP) | |

Title : Reporting and Analysis Plan for: A Two Part Study to Assess i) the Relative Bioavailability and Food Effect of a Novel Tablet Formulation of Boosted-GSK2838232 Compared to Capsule and ii) the Safety and Pharmacokinetics of Repeated Once-Daily Doses of Non boosted GSK2838232

Compound Number : GSK2838232

Effective Date : 07-DEC-2017 (Final 1.0)

#### **Description:**

- The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report for Protocol 205820.
- This RAP is intended to describe the statistical analyses for safety and pharmacokinetic analyses required for the study.
- This RAP will be provided to the study team members to convey the content of the Statistical Analysis Complete (SAC) deliverable.

#### **RAP Authors:**

| Approver | Date | Approval Method |
|---|---|---|
| Principal Biostatistician (PCPS, GSK) | 06-DEC-2017 | e-mail approval |
| PPD | 12-DEC-2017 | e-mail approval |
| Principal Biostatistician (PAREXEL EP Berlin) | | |
| PPD | 12-DEC-2017 | e-mail approval |
| QCD Senior Scientific (PAREXEL Quantitative | | |
| Clinical Development) | | |

Copyright 2017 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

# **RAP Team Approvals:**

| Approver | Date | Approval Method |
|---|---|---|
| PPD | 12-DEC-2017 | e-mail approval |
| Director, Clinical Pharmacology (CPMS, GSK) | | |
| PPD | 12-DEC-2017 | e-mail approval |
| Principal Clinical Research Scientist (CPSSO, | | |
| GSK) | | |
| PPD | 06-DEC-2017 | e-mail approval |
| Sm Executive Medical Director (GSK) | | |
| PPD | 12-DEC-2017 | e-mail approval |
| Principal Programmer (PCPS, GSK) | | |
| PPD | 07-DEC-2017 | e-mail approval |
| Principal Data Manager (CPSSO, GSK) | | |

# **Clinical Statistics and Clinical Programming Line Approvals:**

| Approver | Date | Approval Method |
|-------------------------------------|-------------|-----------------|
| PPD | 07-DEC-2017 | e-mail approval |
| Director, Biostatistics (PCPS, GSK) | | |
| PPD | 12-DEC-2017 | e-mail approval |
| Manager, Programming (PCPS, GSK) | | |

# **TABLE OF CONTENTS**

| | | | | Page |
|---|---|---|---|---|
| DΙV | /ISION | | | 1 |
| 1. | INTRO | ODUCTIC | DN | 6 |
| 2. | SUMN<br>2.1 | | KEY PROTOCOL INFORMATIONs to the Protocol Defined Statistical Analysis Plan | |
| | 2.2<br>2.3 | Study C<br>Study D | bjectives and Endpointsesign | 8 |
| _ | 2.4 | | al Hypotheses/Statistical Analysis | |
| 3. | 9LAN<br>3.1<br>3.2 | Interim A | ALYSESAnalysesalyses | 12 |
| 4. | ANAL<br>4.1 | | PULATIONSI Deviations | |
| 5. | | | ONS FOR DATA ANALYSES AND DATA HANDLING | 14 |
| | 5.1<br>5.2 | Study T | reatment & Sub-group Display Descriptorse Definitions | 14 |
| | 5.3<br>5.4 | | ntre Studiesation of Covariates, Other Strata and Subgroups | |
| | 5.5<br>5.6 | Multiple | Comparisons and Multiplicityonsiderations for Data Analyses and Data Handling | |
| | 0.0 | Conven | tions | 15 |
| 6. | | | _ATION ANALYSES | |
| | 6.1 | | w of Planned Analyses | |
| | 6.2<br>6.3 | Disposit | tion of Participants<br>aphic and Baseline Characteristics | 17<br>17 |
| | 6.4 | | nitant Medications | |
| | 6.5 | | ent Compliance and Protocol Deviations | |
| | 6.6 | | of Exposure | |
| 7. | EFFIC | CACY AN | ALYSES | 18 |
| 8. | | | YSES | |
| | 8.1 | Adverse | Events Analyses | 19 |
| | 8.2 | | Events of Special Interest Analyses | |
| | 8.3<br>8.4 | | Laboratory Analysesafety Analyses | |
| 9. | PHAR | | NETIC ANALYSES | |
| | 9.1 | Primary | Pharmacokinetic Analyses | 20 |
| | | 9.1.1 | Endpoint / Variables | |
| | | | 9.1.1.1 Drug Concentration Measures | |
| | | | 9.1.1.2 Derived Pharmacokinetic Parameters | |
| | | 9.1.2 | Summary Measure | |
| | | 9.1.3 | Population of Interest | 21 |

| 2 | n | $\mathbf{L}$ | О | 2 | r |
|---|---|--------------|---|---|---|
| | u | : ) | n | _ | ı |

| | | 9.1.4<br>9.1.5 | Strategy for Intercurrent (Post-Randomization) Events Statistical Analyses / Methods | 21 |
|---|---|---|---|---|
| | | | Statistical Methodology Specification | |
| | 9.2 | | ary Pharmacokinetic Analyses | |
| | | 9.2.1 | Endpoint / Variables | |
| | | | 9.2.1.1 Drug Concentration Measures | |
| | | | 9.2.1.2 Derived Pharmacokinetic Parameters | |
| | | 9.2.2 | Summary Measure | |
| | | 9.2.3 | Population of Interest | |
| | | 9.2.4 | Strategy for Intercurrent (Post-Randomization) Events | |
| | | 9.2.5 | Statistical Analyses / Methods | |
| | 0.0 | | Statistical Methodology Specification | 26 |
| | 9.3 | Explorat | ory Pharmacokinetic Analyses | 28 |
| 10. | POPU | LATION F | PHARMACOKINETIC (POPPK) ANALYSES | 28 |
| 11. | PHAR | MACODY | NAMIC ANALYSES | 28 |
| 12. | PHAR | MACOKIN | NETIC / PHARMACODYNAMIC ANALYSES | 28 |
| 10 | DEEE | DENCES | | 20 |
| 13. | KEFEI | KENCES. | | ∠0 |
| 14. | APPEI | NDICES | | 28 |
| | 14.1 | Appendi | x 1: Protocol Deviation Management and Definitions for Per | |
| | | Protocol | Population | |
| | 14.2.1 | Exclusio | ns from Per Protocol Population | 28 |
| | 14.2 | Appendi | x 2: Schedule of Activities | 29 |
| | 14.2.1 | Protocol | Defined Schedule of Events | 29 |
| | | | Schedule of Assessments for Part 1A and Part 1B: Single | |
| | | | Dose RBA ± Food | 29 |
| | | | Schedule of Assessments for Part 2: Repeated Doses for | |
| | | | 11 days: | 31 |
| | 14.3 | | x 3: Assessment Windows | |
| | 14.3.1 | Definition | ns of Assessment Windows for Analyses | 34 |
| | 14.4 | Appendi | x 4: Study Phases and Treatment Emergent Adverse | |
| | | Events | | 35 |
| | 14.4.1 | Study Ph | nases | |
| | | | 14.4.4.1 Study Phases for Concomitant Medication | |
| | 14.4.2 | Treatme | nt Emergent Flag for Adverse Events | 35 |
| | | | Events Assignment to Treatment Period for Part 1 | |
| | 14.4.4 | | itant Medication Assignment to Treatment Period for Part 1 | |
| | 14.5 | | x 5: Data Display Standards & Handling Conventions | |
| | 14.5.1 | Reportin | g Process | 37 |
| | | | g Standards | |
| | 14.5.3 | | g Standards for Pharmacokinetic Data | |
| | 14.6 | | x 6: Derived and Transformed Data | |
| | | | opulation | |
| | 14.6.4 | Safety | | 41 |
| | | | cokinetic | |
| | 14.6.6 | Population | on Pharmacokinetic (PopPK) | 42 |

| 205820 |
|----------|
| ・ソハトな・ソハ |

| 14.6.7 Pharmac | odynamic | .42 |
|-------------------|--------------------------------------------------|-----|
| | 7. Reporting Standards for Missing Data | |
| | e Withdrawals | |
| | of Missing Data | |
| | of Missing and Partial Dates | |
| 14.8 Appendix | 8: Values of Potential Clinical Importance | .45 |
| | ry Values | |
| 14.8.2 ECG | * | .46 |
| 14.8.3 Vital Sign | ns | .46 |
| 14.9 Appendix | 9: Population Pharmacokinetic (PopPK) Analyses | .47 |
| 14.9.1 Population | on Pharmacokinetic (PopPK) Dataset Specification | .47 |
| 14.9.2 Population | n Pharmacokinetic (PopPK) Methodology | .47 |
| 14.10 Appendix | 10: Pharmacokinetic / Pharmacodynamic Analyses | .48 |
| 14.10.1 | Pharmacokinetic / Pharmacodynamic Dataset | |
| Specifica | tion | .48 |
| 14.10.2 | Pharmacokinetic / Pharmacodynamic Methodology | .48 |
| 14.11 Appendix | 11: Abbreviations & Trade Marks | .49 |
| 14.11.1 | Abbreviations | .49 |
| 14.11.2 | Trademarks | .51 |
| 14.12 Appendix | c 12: List of Data Displays | .52 |
| 14.12.1 | Data Display Numbering | .52 |
| 14.12.2 | Mock Example Shell Referencing | .52 |
| 14.12.3 | Deliverable [Priority] | .52 |
| 14.12.4 | Study Population Tables | .53 |
| 14.12.5 | Efficacy Tables | |
| 14.12.6 | Efficacy Figures | .56 |
| 14.12.7 | Safety Tables | .57 |
| 14.12.8 | Safety Figures | .62 |
| 14.12.9 | Pharmacokinetic Tables | .63 |
| 14.12.10 | Pharmacokinetic Figures | .65 |
| 14.12.11 | Pharmacokinetic Population (PopPK) Tables | |
| 14.12.12 | Pharmacokinetic Population (PopPK) Figures | |
| 14.12.13 | Pharmacodynamic Tables | .67 |
| 14.12.14 | Pharmacodynamic Figures | .67 |
| 14.12.15 | Pharmacokinetic / Pharmacodynamic Tables | |
| 14.12.16 | Pharmacokinetic / Pharmacodynamic figures | .67 |
| 14.12.17 | ICH Listings | .68 |
| 14.12.18 | Non-ICH Listings | .74 |
| 14.13 Appendix | 13: Example Mock Shells for Data Displays | .75 |

## 1. INTRODUCTION

The purpose of this reporting and analysis plan (RAP) is to describe the analyses to be included in the Clinical Study Report for Protocol:

| Revision Chronology | y: | |
|---|---|---|
| 2017N322544_00 | 09-JUN-2017 | Original |
| 2017N322544_01 | 17-JUL-2017 | Amendment No.: 1. |
| | | The protocol was amended to include an assessment of neuropsychiatric adverse events at each AE enquiry as well as a statement to inform FDA of any grade 2 or higher alteration in personality-behavior or in mood or altered mental status within 7 days, per FDA request. |
| | | Minor typographical errors were also amended in the Schedule of Assessments, the Exclusion Criteria and the Study Assessment and Procedures. |

# 2. SUMMARY OF KEY PROTOCOL INFORMATION

# 2.1 Changes to the Protocol Defined Statistical Analysis Plan

There were no changes or deviations to the originally planned statistical analysis specified in the amended protocol (dated: 17-JUL-2017).

# 2.2 Study Objectives and Endpoints

Part 1.

| Objectives | Endpoints |
|---|---|
| Primary Objectives | Primary Endpoints |
| To assess the relative bioavailability of a<br>novel GSK2838232 tablet formulations<br>versus the capsule formulation (Part 1A) | AUC(0-∞) and Cmax |
| To assess the effect of food on<br>GSK2838232 exposure of the tablet<br>formulation (Part 1A and Part 1B) | AUC(0-∞), Cmax, and tmax |
| Secondary Objectives | Secondary Endpoints |
| To investigate the safety and tolerability of<br>GSK2838232 following single dose<br>administration as tablets or capsules, with<br>Ritonavir (RTV) | GSK2838232 safety parameters: adverse events (AEs); absolute values and changes over time of clinical laboratory evaluations (hematology, clinical chemistry, urinalysis), vital signs, and 12-lead electrocardiogram (ECG) parameters from pre-dose values |
| To characterize the pharmacokinetics (PK) of GSK2838232 after administration of a novel tablet formulation and capsule formulation with food, and the tablet formulation given without food | • tlag, tmax, t½, tlast, C24, and AUC(0-t) |

Part 2.

| Objectives | Endpoints |
|---|---|
| Primary Objectives | Primary Endpoints |
| To assess the safety of GSK2838232<br>administered as non-boosted once-daily<br>doses of a tablet formulation for 11 days | <ul> <li>GSK2838232 safety parameters: AEs; absolute values<br/>and changes over time of clinical laboratory<br/>evaluations (hematology, clinical chemistry, urinalysis),<br/>vital signs, and ECG parameters from pre-dose values</li> </ul> |
| To assess the PK of GSK2838232<br>administered as non-boosted once-daily<br>doses of a tablet formulation for 11 days | <ul> <li>Day 1 dose: AUC(0-τ), Cmax, Cτ, tmax, tlag</li> <li>Day 11 dose: AUC(0-τ), AUC(0-∞), Cmax, Cτ, tmax, t½, tlast</li> </ul> |
| Secondary Objectives | Secondary Endpoints |
| To assess time to steady-state of<br>GSK2838232 when administered as non-<br>boosted once-daily doses of a tablet<br>formulation for 11 days | Pre-dose concentrations on Days 2 to 11 |
| To assess accumulation of GSK2838232<br>when administered as non-boosted once-<br>daily doses of a tablet formulation for 11<br>days | <ul> <li>Accumulation ratios: Ro[AUC(0-τ)], R(Cmax), R(Cτ)</li> </ul> |

AUC( $0-\tau$ ) = Area under the curve (Area under the plasma drug concentration-time curve from pre-dose to the end of the dosing interval); AUC( $0-\infty$ ) = Area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time; Cmax = Maximum observed concentration; C $\tau$ =Observed concentration at the end of the dosing interval;  $t\frac{1}{2}$  = Apparent terminal phase half-life; tmax = Time of occurrence of Cmax; tlag = Lag time (time delay between drug administration and first observed concentration above LOQ in plasma); AUC(0-t) = Area under the concentration-time curve from zero up to last quantifiable concentration; tlast = Time of last quantifiable concentration

## 2.3 Study Design

#### **Overview of Study Design and Key Features**

This study is divided into two study parts, Part 1 (Table 1 and Figure 1) and Part 2 (Figure 2).

Table 1 Study Design for Part 1

| Sequence | N | Part 1A | | Part 1B |
|----------|---|----------|----------|----------|
| Coquence | | Period 1 | Period 2 | Period 3 |
| 1 | 6 | А | В | С |
| 2 | 6 | В | A | |

- All treatments in Part 1A to be administered with RTV in fed state, following two RTV pre-doses.
- 2. There will be a washout of at least 10 days between each Period.
- 3. Treatment A =  $GSK2838232\ 200\ mg/r$  (as  $4\times 50\ mg$ ) capsule formulation, fed, normal fat (i.e., approximately 30%) meal (reference).
- 4. Treatment B = GSK2838232 200 mg/r (as 2 x 100 mg) tablet formulation, fed, normal fat (i.e., approximately 30%) meal.
- 5. Treatment C = GSK2838232 200 mg/r (as 2 x 100 mg) tablet, confirmed from Part 1A, fasted.

Figure 1 Part 1: Single Dose, Food Effect Study Design Schematic



Treatments A and B will be Capsule and Tablet administered in a randomized crossover design with 100 mg Ritonavir with food (fed state) (Part 1A).

Treatment C will be Tablet assessed in Part 1A, administered with 100 mg Ritonavir without food (fasted state) (Part 1B)



#### **Design Features**

#### Part 1:

- Part 1 is a relative bioavailability study (Table 1) that will further subdivide into two parts (Part 1A and Part 1B).
- In Part 1A, the safety and PK of a novel tablet formulation of GSK2838232 will be evaluated in open label, randomized, cross over fashion against the capsule formulation as reference.
- Each actual treatment dose will be separated by a minimum 10 day washout period. Part 1A will be studied in the fed state using a normal fat (i.e., approximately 30%) meal in all participants.
- The safety and PK will be evaluated, and the tablet will be evaluated for suitability, and further clinical assessment in Part 1B, where the tablet will be administered in the fasted state to understand the impact of food on relative bioavailability.
- GSK2838232 as tablets or capsules (at a 200 mg dose level) will be administered with 100 mg RTV, after two pre-doses of 100 mg RTV once daily (QD) over 48 h. The use of RTV priming is an aspect of GSK2838232 clinical development (specifically relative bioavailability studies) so far and allows a more accurate assessment of what will ultimately happen in the repeat-dose clinical studies with GSK2838232 when boosted with RTV. In Part 2 of the study, however, GSK2838232 will be administered unboosted and no RTV will be co administered.
- Participants will have a screening visit within 30 days prior to first dose, a
  minimum 10-day washout period between doses, and a follow-up visit 7 to 14
  days after the last dose. The maximum duration of study participation will be
  approximately 9 to 10 weeks.

After completion of Part 1A, preliminary PK data will be analyzed, and a decision will be made based on tolerability, relative bioavailability PK criteria, as well as feasibility considerations, as to whether the tablet formulation will be used to conduct Part 1B (fasted) and Part 2.

#### Part 2:

Part 2 will evaluate non-RTV boosted GSK2838232, given as single daily doses

| Overview of Study | Design and Key Features |
|---|---|
| | <ul> <li>for 11 days in a separate cohort of participants (N=8; 6A/2P).</li> <li>The placebo tablet supplied will not be identical to GSK2838232 and as such will be administered by site staff via an opaque card/paper tube to facilitate the single blind (i.e., the Principal Investigator [PI] and the participants themselves will be blinded as to their treatment).</li> <li>The dose chosen for Part 2 will depend upon the preliminary results of the tablet in Part 1A but is likely to be, but will not exceed, 500 mg (i.e., 5 x 100 mg tablets) QD.</li> <li>Participants will have a screening visit within 30 days prior to first dose, and a follow-up visit 7 to 14 days after the last dose. The maximum duration of study participation will be approximately 8 to 9 weeks.</li> <li>Details of the assessments and procedures participants will undergo are listed in Section 9 of the Clinical Study Protocol (CSP). The time points and visits are provided in the schedule of assessments, (Table 2 and Table 3 of the CSP for the Schedule of assessments for study Parts 1 and 2 respectively).</li> </ul> |
| Treatment Assignment | <ul> <li>The dose for Part 1A and Part 1B of this study will be 200 mg (achieved as either 4 x 50 mg capsules or 2 x 100 mg tablets) administered with 100 mg RTV.</li> <li>The dose for Part 2 will be confirmed from Part 1A but is likely to be, and will not exceed, 500 mg (as 5 x 100 mg tablets).</li> <li>The randomization number will determine the allocation of treatment sequences (ABC or BAC) for Part 1, and of treatment (GSK2838232 without RTV or placebo) for Part 2.</li> <li>Part 1 treatments: <ul> <li>Treatment A = GSK2838232 200 mg/r (as 4 x 50 mg) capsule formulation, fed, normal fat (i.e., approximately 30%) meal (reference).</li> <li>Treatment B = GSK2838232 200 mg/r (as 2 x 100 mg) tablet formulation, fed, normal fat (i.e., approximately 30%) meal.</li> <li>Treatment C = GSK2838232 200 mg/r (as 2 x 100 mg) tablet, formulation confirmed from Part 1A, fasted.</li> </ul> </li> <li>Part 2 treatments: <ul> <li>Treatment D = GSK2838232 500 mg/r (as 5 x 100 mg) tablet formulation, fed, normal fat (i.e., approximately 30%) meal (reference).</li> <li>Treatment E = Placebo</li> </ul> </li> <li>The dose chosen for Part 2 will depend upon the preliminary results of the tablet in Part 1A but is likely to be, but will not exceed, 500 mg (i.e., 5 x 100 mg tablets) QD.</li> </ul> |
| Interim Analysis | No formal interim analyses are planned for this study; an informal analysis of data from Part 1A of the study will decide the dose and formulation to be administered in Part 1B and Part 2. |

## 2.4 Statistical Hypotheses/Statistical Analysis

No formal statistical hypotheses will be tested. Analysis will be descriptive and exploratory. An estimation approach providing point estimates and corresponding confidence intervals will be used, where appropriate.

#### Part 1A Relative Bioavailability

Part 1A of this study is designed to estimate the bioavailability of a novel GSK2838232 tablet formulations versus the capsule formulation at 200 mg/r. No formal hypothesis will be tested. The dependent variable will be the log-transformed PK parameters of interest (AUC(0-∞) and Cmax) and the independent variables will include fixed effects for treatment (table or capsule), sequence and period, and participant (sequence) as a random effect. For each primary pharmacokinetic endpoint, point estimates and corresponding 90% confidence intervals will be constructed for the ratio of the geometric mean of the test treatment (GSK2838232 200 mg/r tablet) to the geometric mean of the reference treatment (GSK2838232 200 mg/r capsule), μ(test)/μ(reference).

#### Part 1A and 1B Food Effect

Part 1A and 1B of this study are designed to evaluate the effect of food on GSK2838232 exposure of the tablet formulation. No formal hypothesis will be tested. The dependent variable will be the log-transformed PK parameters of interest (AUC( $0-\infty$ ) and Cmax) and the independent variables will include a fixed effect for treatment (with or without food) and participant as a random effect. The estimated difference and confidence interval (CI) obtained on the log scale will be exponentiated to provide an estimate of the fed to fasted ratio and its associated 90% CI.

For the parameter tmax the corresponding non-parametric analysis will be performed on the original scale using CIs for the estimation of the treatment difference based on the Hodges-Lehman estimator.

#### **Part 2 Steady State Assessments**

Part 2 of this study is designed to assess time to steady-state of GSK2838232 when administered as non-boosted once-daily doses of a tablet formulation for 11 days. No formal hypothesis will be tested. Mean plasma GSK2838232 pre-dose values between Days 2 through 11 and  $C\tau$  of Day 11 will be plotted against time. Achievement of plasma GSK2838232 steady-state will be assessed by calculating the 90% CI of the slope of the linear regression of log  $(C\tau)$  versus time. The dependent variable in the linear regression model will be log  $(C\tau)$  and the model will include a random intercept effect for participant and a fixed slope effect for study day. Steady state will be reached if the 90% CI for the slope estimate includes zero.

#### Part 2 Accumulation

Part 2 of this study is designed to assess accumulation of GSK2838232 when administered as non-boosted once-daily doses of a tablet formulation for 11 days. No formal hypothesis will be tested. The extent of accumulation of GSK2838232 will be

evaluated by comparing AUC(0- $\tau$ ), Cmax and C $\tau$  between Day 11 and Day 1. For each of these comparisons an analysis of variance will be conducted on the log scale. The difference between Day 11 and Day 1 least square (LS) means and a 90% CI will be computed by fitting a mixed effects model with the log-transformed PK parameter as the dependent variable, day as a fixed effect and participant as a random effect. The estimated difference and confidence interval obtained on the log-scale will be exponentiated to provide an estimate of the Day 11 to Day 1 ratio and its associated 90% CI. If the model fails to converge, participants will be fit as a fixed effect.

#### 3. PLANNED ANALYSES

# 3.1 Interim Analyses

No formal interim analyses are planned for this study. The dose and formulation to be administered in Part 1B and Part 2 will be decided, based on the outcome and results of an informal analysis of preliminary safety and PK data from Part 1A of the study. In addition, and descriptive analysis of preliminary safety and PK data from Part 1 and 2 of the study will be performed.

### 3.2 Final Analyses

The final planned primary analyses will be performed after the completion of the following sequential steps:

- o All participants have completed the study as defined in the protocol.
- All required database cleaning activities have been completed and final database release and database freeze has been declared by Data Management.
- o All criteria for unblinding the randomisation codes have been met.
- o Randomisation codes have been distributed according to PAREXEL procedures.

#### 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| Screened | All participants who were screened for eligibility | <ul> <li>Study Population</li> </ul> |
| Safety | <ul> <li>The Safety Population will include all participants who received at least 1 dose of the study treatment (including placebo) with at least 1 post-baseline safety assessment.</li> <li>This population will be based on the treatment the participant received.</li> <li>The population will be defined separately for Part 1 and Part 2 of the study.</li> </ul> | Safety and Demography |

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| PK | <ul> <li>All participants in the Safety population who had at least 1 non-missing PK assessment (Non-quantifiable [NQ] values will be considered as non-missing values). Pharmacokinetic samples that may be affected by protocol deviations will be reviewed by the study team to determine whether the sample will be excluded.</li> <li>This population will be based on the treatment the participant received.</li> <li>The population will be defined separately for Part 1A, Part 1B and Part 2 of the study.</li> </ul> | • PK |

#### NOTES:

 Please refer to Appendix 8: List of Data Displays which details the population to be used for each displays being generated.

#### 4.1 Protocol Deviations

Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, participant management or participant assessment) will be summarised and listed.

Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan (PDMP) version final 1.0 dated 22 Aug 2017.

- Data will be reviewed prior to freezing the database to ensure all important deviations are captured and categorised on the protocol deviations dataset.
- This dataset will be the basis for the summaries and listings of protocol deviations.

A separate summary and listing of all inclusion/exclusion criteria deviations will also be provided. This summary will be based on data as recorded on the inclusion/exclusion page of the Electronic Case Record Form (eCRF).

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

# 5.1 Study Treatment & Sub-group Display Descriptors

| | Treatment Group Descriptions – Part 1 | | |
|---|---|---|---|
| | RandAll NG | Data Displays for Reporting | |
| Code | Description | Description | Order in TFL |
| C1 | GSK2838232 200 mg/r (as 4 x 50 mg) capsule formulation, fed, normal fat (i.e., approximately 30%) meal (reference) | GSK 200 mg/r capsule fed | 1 |
| T1 | GSK2838232 200 mg/r (as 2 x 100 mg) tablet formulation, fed, normal fat (i.e., approximately 30%) meal | GSK 200 mg/r tablet fed | 2 |
| T2 | GSK2838232 200 mg/r (as 2 x 100 mg) tablet, confirmed from Part 1A, fasted | GSK 200 mg/r tablet fasted | 3 |

Treatment comparisons will be displayed as follows using the descriptors as specified:

- 1. GSK 200 mg/r tablet fed vs GSK 200 mg/r capsule fed
- 2. GSK 200 mg/r tablet fed vs GSK 200 mg/r tablet fasted

| | Treatment Group Descriptions – Part 2 | | |
|---|---|---|---|
| RandAll NG Data Displays for Reporting | | ıg | |
| Code | Description | Description | Order in TFL |
| T3 | GSK2838232 500 mg/r (as 5 x 100 mg) tablet formulation, fed, normal fat (i.e., approximately 30%) meal (reference). | GSK 500 mg/r tablet fed | 2 |
| Р | Placebo | Placebo | 1 |

Treatment comparisons will be displayed as follows using the descriptors as specified:

1. GSK 500 mg/r tablet fed vs Placebo

#### 5.2 Baseline Definitions

For all endpoints (except as noted in baseline definitions) the baseline value will be the latest pre-dose assessment, including those from unscheduled visits. If time is not collected, Day 1 assessments are assumed to be taken prior to first dose and used as baseline. In part 1, baseline definitions are applicable to each period.

| Parameter | Study Assessments Considered As Baseline | | | | Baseline Used in |
|---|---|---|---|---|---|
| | Screening | Day -2 | Day -1 | Day 1 (Pre-Dose) | Data Display |
| Safety Data | | • | | • | |
| Vital Signs | X | X* | X | X | Mean of replicate assessments on Day |
| ECG | Х | X* | Х | X | Mean of replicate assessments on Day |
| Laboratory tests | Х | X* | Х | | Day -1 |

<sup>\*</sup> Vital Sign, ECG and laboratory tests are not collected at day -2 for Part 2.

Unless otherwise stated, if baseline data is missing no derivation will be performed and baseline will be set to missing.

#### 5.3 Multicentre Studies

Not applicable.

# 5.4 Examination of Covariates, Other Strata and Subgroups

Not applicable.

# 5.5 Multiple Comparisons and Multiplicity

Not applicable.

# 5.6 Other Considerations for Data Analyses and Data Handling Conventions

Other considerations for data analyses and data handling conventions are outlined in the appendices:

| Section | Component |
|---------|----------------------------------------------------------------|
| 14.3 | Appendix 3: Assessment Windows |
| 14.4 | Appendix 4: Study Phases and Treatment Emergent Adverse Events |
| 14.5 | Appendix 5: Data Display Standards & Handling Conventions |
| 14.6 | Appendix 6: Derived and Transformed Data |
| 14.7 | Appendix 7: Reporting Standards for Missing Data |

| Section | Component |
|---------|-----------------------------------------------------|
| 14.8 | Appendix 8: Values of Potential Clinical Importance |

#### 6. STUDY POPULATION ANALYSES

## 6.1 Overview of Planned Analyses

The study population analyses will be based on the Safety Population, unless otherwise specified.

Study population analyses including analyses of participant's disposition, protocol deviations, demographic and baseline characteristics, prior and concomitant medications, and exposure and treatment compliance will be based on GSK Core Data Standards. Details of the planned displays are presented in Appendix 12: List of Data Displays.

## 6.2 Disposition of Participants

A summary of the number of participants in each of the analysis populations described in Section 4 will be provided and this table will be displayed by treatment/sequence and overall of each part. A listing of participants excluded from analysis populations will also be provided.

A summary of participant status and reason for study withdrawal will be provided. This display will show the number and percentage of participants who withdrew from the study, including primary reasons for study withdrawal.

A summary of study treatment status will be provided. This display will show the number and percentage of participants who have completed the study or have discontinued study treatment and a summary of the primary reasons for discontinuation of study treatment. A listing of study treatment discontinuation will be generated. The listing will include last dose date, and reasons for study treatment discontinuation as well as study part and period, when applicable, of discontinuation.

# 6.3 Demographic and Baseline Characteristics

The demographic characteristics (e.g., age, ethnicity, sex, height, and body weight) will be summarized and listed by participant. Race will be summarized and listed separately from the other demographic characteristics. Age, height, body mass index (BMI) and weight will be summarized using the mean, standard deviation, minimum, median, and maximum. The count and percentage will be computed for sex, race and ethnicity. The summary table will be displayed by treatment/treatment sequence and overall of each part.

Medical conditions present at screening will be summarized by treatment/treatment sequence and overall of each part, and listed by participant.

Substance use will be listed.

#### 6.4 Concomitant Medications

Concomitant medications will be coded using GSK Drug coding dictionary, summarized by treatment and study part, and listed by participant. The summary of concomitant

medications will show the number and percentage of participants taking concomitant medications by ingredient. Multi-ingredient products will be summarized by their separate ingredients rather than as a combination of ingredients. Anatomical Therapeutic Chemical (ATC) classification Level 1 (Body System) information will be included in the dataset created, however, will not appear on the listing or summary.

In the summary of concomitant medications, each participant is counted once within each unique ingredient. For example, if a participant takes amoxicillin on two separate occasions, the participant is counted only once under the ingredient "amoxicillin".

In the summary of concomitant medications, the ingredients will be summarized by the base only, using CMBASECD and CMBASE.

# 6.5 Treatment Compliance and Protocol Deviations

Information of each participant not received the correct treatment during each treatment period, the reason for not receiving the correct treatment, and any other protocol deviations will be summarized by treatment /sequence and overall of each part, and listed by participant and period (treatment). In addition, a listing will be provided including dose administered along with dosing dates and time for the investigational product.

Participants who did not satisfy all inclusion and exclusion criteria and corresponding criteria that were violated will be summarized and listed.

For the food effect of Part 1, a by-participant listing of the meal data will also be generated including start and stop date and time of meal, dosing time, type of meal and whether the totality of the meal was ingested.

### 6.6 Extent of Exposure

A by-participant summary of treatments administered in each part will be generated, with dose, and dosing start date, dosing end date and number of dose. A by-participant listing of data on participant exposure will be generated including dose date and time, unit, formulation, route and frequency.

#### 7. EFFICACY ANALYSES

Not applicable.

## 8. SAFETY ANALYSES

The safety analyses will be based on the "Safety Population", unless otherwise specified.

## 8.1 Adverse Events Analyses

Adverse events analyses including the analysis of adverse events (AEs), Serious (SAEs) and other significant AEs will be based on GSK Core Data Standards. The details of the planned displays are provided in Appendix 12: List of Data Displays.

## 8.2 Adverse Events of Special Interest Analyses

Not applicable.

## 8.3 Clinical Laboratory Analyses

Laboratory evaluations including the analyses of Chemistry laboratory tests, Hematology laboratory tests, Urinalysis, and liver function tests will be based on GSK Core Data Standards. The details of the planned displays are in Appendix 12: List of Data Displays.

## 8.4 Other Safety Analyses

The analyses of non-laboratory safety test results including ECGs and vital signs will be based on GSK Core Data Standards, unless otherwise specified. The details of the planned displays are presented in Appendix 12: List of Data Displays.

#### 9. PHARMACOKINETIC ANALYSES

## 9.1 Primary Pharmacokinetic Analyses

#### 9.1.1 Endpoint / Variables

### 9.1.1.1 Drug Concentration Measures

Pharmacokinetic data will be presented in graphical and/or tabular form and will be summarized descriptively. Plasma GSK2838232 concentration-time data will be listed by participant, treatment group and time and summarized by treatment group and time for each part of the study. Individual participant profiles for GSK2838232 concentration-time data will be presented on both a linear and semi-log scale. Linear and semi-log figures for mean and median GSK2838232 plasma concentrations versus time will also be generated.

Refer to Appendix 5: Data Display Standards & Handling Conventions (Section 14.5.3 Reporting Standards for Pharmacokinetic).

#### 9.1.1.2 Derived Pharmacokinetic Parameters

Pharmacokinetic parameters will be calculated by standard non-compartmental analysis according to current working practices and using the currently supported version of WinNonlin. All calculations of non-compartmental parameters will be based on actual sampling times. Pharmacokinetic parameters listed will be determined from the plasma concentration-time data, as data permits.

#### Part 1:

| Parameter | Parameter Description |
|---|---|
| AUC(0-∞) | Area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time will be calculated as: |
| | AUC = AUC(0-last) + C(last) / lambda_z |
| Cmax | Maximum observed concentration, determined directly from the concentration-time data |
| tmax | Time of occurrence of Cmax, determined directly from the concentration-time data |

Part 2

| Parameter | Parameter Description |
|---|---|
| AUC(0-τ) | Area under the plasma drug concentration-time curve from pre-dose to the end of the dosing interval (where $\tau$ = 24 h) (Day 1 and Day 11) |
| AUC(0-∞) | Area under the concentration-time curve extrapolated to infinity will be calculated as: AUC = AUC(0-last) + C(last) / lambda_z |
| Cmax | Maximum observed concentration, determined directly from the concentration-time data. (Day 1 and Day 11) |
| tmax | Time of occurrence of Cmax, determined directly from the concentration-time data (Day 1 and Day 11) |
| tlag | Lag-time (time delay between drug administration and first observed concentration), |

| Parameter | Parameter Description |
|---|---|
| | determined directly from the concentration-time data (Day 1) |
| tlast | Time of last quantifiable concentration, determined directly from the concentration-time data (Day 11) |
| t½ | Apparent terminal phase half-life, calculated as; t½ = ln2 / lambda_z (Day 11) |
| Сτ | Observed concentration at the end of the dosing interval, determined directly from the concentration-time data (where $\tau$ = 24 h) (Day 1 and Day 11) |
| Ctrough | Observed pre-dose concentrations on Days 2 to 11, determined directly from the concentration-time data |

#### NOTES:

 C24, Cτ and Ctrough will be extracted from the concentration data by Clinical Statistics group and merged with other calculated PK parameters provided by CPMS.

All the derived parameters described above will be listed. For each of these parameters, except tmax and tlag, the following summary statistics will be calculated for each treatment group: n, arithmetic mean, standard deviation (SD), median, minimum, maximum, geometric mean with associated 90% CI, standard deviation of logarithmically transformed data, and the between-participant CV (%CVb) based on the geometric mean for the loge-transformed PK parameters. For tmax and tlag, median, maximum, minimum, arithmetic mean and standard deviation will be calculated.

#### 9.1.2 Summary Measure

The measures used for the treatment comparisons are the following:

- For part 1;  $AUC(0-\infty)$ , Cmax, and, for food effect, tmax.
- For part 2; Not applicable.

## 9.1.3 Population of Interest

The primary pharmacokinetic analyses will be based on the Pharmacokinetic population, unless otherwise specified.

### 9.1.4 Strategy for Intercurrent (Post-Randomization) Events

Not applicable.

#### 9.1.5 Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 12: List of Data Displays and will be based on GSK Data Standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 9.1.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

#### Statistical Methodology Specification

The following pharmacokinetic statistical analyses will only be performed if sufficient data is available (i.e. if participants have well defined plasma profiles).

#### Part 1A Relative Bioavailability

#### **Endpoint / Variables**

AUC(0-∞) and Cmax

#### **Model Specification**

AUC(0-∞) and Cmax will be separately analysed using a mixed effects model. The dependent variable will be the log-transformed PK parameters of interest (AUC(0-∞) and Cmax) and the independent variables will include fixed effects for treatment (GSK2838232 200 mg/r tablet or GSK2838232 200 mg/r capsule), sequence and period, and participant (sequence) as a random effect.

## **Model Checking & Diagnostics**

- Model assumptions will be applied, but appropriate adjustments may be made based on the data.
- The Kenward and Roger method for approximating the denominator degrees of freedom and correcting for bias in the estimated variance-covariance of the fixed effects will be used.
- Normality assumptions underlying the model used for analysis will be examined by obtaining a
  normal probability plot of the residuals and a plot of the residuals versus the fitted values (i.e.
  checking the normality assumption and constant variance assumption of the model
  respectively) to gain confidence that the model assumptions are reasonable.
- If there are any departures from the distributional assumptions, alternative models will be explored using appropriate transformed data.

#### **Model Results Presentation**

- Geometric least-squares means for each treatment (tablet or capsule), point estimates and associated 90% confidence intervals for the ratios for each parameter will be produced in tabular format. Estimates of within-subject variability (%CVw) will also be provided. %CVw represents a pooled measure of within-subject variability across all treatments.
- Comparative plots of individual PK parameters will be generated by treatment on linear and semi-logarithmic scales.
- Plots of adjusted geometric mean ratio of test to reference treatment together with 90% confidence intervals will be produced.
- Listing of individual PK parameter ratios will be generated.
- Supportive SAS output from statistical analysis will be generated.

#### **Subgroup Analyses**

Not applicable

#### **Sensitivity and Supportive Analyses**

Not applicable

#### Part 1 A and 1B Food Effect

#### **Endpoint / Variables**

AUC(0-∞) and Cmax

#### **Model Specification**

- AUC(0-∞) and Cmax will be separately analysed using a mixed effects model. The dependent variable will be the log-transformed PK parameters of interest (AUC(0-∞) and Cmax) and the independent variables will include a fixed effect for treatment (with or without food) and participant as a random effect.
- To assess the effect of food on GSK2838232 exposure of the tablet formulation (Part 1A and Part 1B)

#### **Model Checking & Diagnostics**

- Model assumptions will be applied, but appropriate adjustments may be made based on the data.
- The Kenward and Roger method for approximating the denominator degrees of freedom and correcting for bias in the estimated variance-covariance of the fixed effects will be used.
- Normality assumptions underlying the model used for analysis will be examined by obtaining a
  normal probability plot of the residuals and a plot of the residuals versus the fitted values (i.e.
  checking the normality assumption and constant variance assumption of the model
  respectively) to gain confidence that the model assumptions are reasonable. If there are any
  departures from the distributional assumptions, alternative models will be explored using
  appropriate transformed data.

#### **Model Results Presentation**

- The estimated difference and CI obtained on the log scale will be exponentiated to provide an
  estimate of the fed to fasted ratio and its associated 90% CI. Estimates of within-subject
  variability (%CVw) will also be provided. %CVw represents a pooled measure of within-subject
  variability across all treatments.
- Comparative plots of individual PK parameters will be generated by treatment on linear and semi-logarithmic scales.
- Plots of adjusted geometric mean ratio of test to reference treatment together with 90% confidence intervals will be produced.
- Listing of individual PK parameter ratios will be generated.
- Supportive SAS output from statistical analysis will be generated.

#### Subgroup Analyses

Not applicable

#### Sensitivity and Supportive Analyses

Not applicable

#### **Endpoint / Variables**

tmax

#### **Model Specification**

- Non-parametric analysis, using PROC NPAR1WAY will be performed on the original scale PK parameters of interest (tmax). The dependent variable will be the original scale PK parameter of interest (tmax) and the independent variables will be treatment (with or without food).
- SAS code:

```
PROC NPAR1WAY data= data hl ALPHA=0.1;
```

CLASS treatment:

VAR pk:

EXACT hl;

/\* where PK parameter pk = tmax\*/

ods select HodgesLehmann;

RUN:

#### Model Checking & Diagnostics

 Model assumptions will be applied, but appropriate adjustments may be made based on the data.

#### **Model Results Presentation**

 90% CIs for the estimation of the treatment difference based on the Hodges-Lehman estimator will be produced

#### **Subgroup Analyses**

Not applicable

#### Sensitivity and Supportive Analyses

Not applicable

# 9.2 Secondary Pharmacokinetic Analyses

#### 9.2.1 Endpoint / Variables

#### 9.2.1.1 Drug Concentration Measures

Refer to Appendix 5: Data Display Standards & Handling Conventions (Section 14.5.3 Reporting Standards for Pharmacokinetic)

#### 9.2.1.2 Derived Pharmacokinetic Parameters

Pharmacokinetic parameters will be calculated by standard non-compartmental analysis according to current working practices and using the currently supported version of WinNonlin. All calculations of non-compartmental parameters will be based on actual sampling times. Pharmacokinetic parameters listed will be determined from the plasma concentration-time data, as data permits.

#### Part 1:

| Parameter | Parameter Description |
|---|---|
| AUC(0-t) | Area under the concentration-time curve from zero up to the last quantifiable concentration will be calculated using the linear trapezoidal rule for each incremental trapezoid and the log trapezoidal rule for each decremental trapezoid |
| tmax | Time to reach Cmax, determined directly from the concentration-time data. |
| tlag | Lag-time (time delay between drug administration and first observed concentration) |
| t½ | Apparent terminal half-life will be calculated as: t½ = ln2 / lambda_z |
| tlast | Time of last quantifiable concentration, determined directly from the concentration-time data. |
| C24 | Observed concentration 24 hours post-dose, determined directly from the concentration-time data. |

#### NOTES:

- Additional parameters may be included as required.
- Lambda\_z is the terminal phase rate constant.

#### Part 2

| Parameter | Parameter Description |
|---|---|
| Ctrough | Observed pre-dose concentrations on Days 2 to 11, determined directly from the concentration-time data |
| Ro[AUC(0-τ)] | Accumulation ratio based on AUC(0- $\tau$ ), determined by; Day 11 AUC(0- $\tau$ ) / Day 1 AUC(0- $\tau$ ) |
| R(Cmax) | Accumulation ratio based on Cmax, determined by; Day 11 Cmax / Day 1 Cmax |
| R(Cτ) | Accumulation ratio based on $C\tau,$ determined by; Day 11 $C\tau$ / Day 1 $C\tau$ |

#### NOTES:

- Additional parameters may be included as required.
- Cτ, and Ctrough will be extracted from the concentration data by Clinical Statistics group and merged with other calculated PK parameters provided by CPMS.

All the derived parameters described above will be listed. For each of these parameters, except tmax and tlag, the following summary statistics will be calculated for each treatment group: n, arithmetic mean, standard deviation (SD), median, minimum, maximum, geometric mean with associated 90% CI, standard deviation of logarithmically transformed data, and the between-participant CV (%CVb) based on the geometric mean for the loge-transformed PK parameters. For tmax and tlag, median, maximum, minimum, arithmetic mean and standard deviation will be calculated.

#### 9.2.2 Summary Measure

The measures used for the treatment comparisons are the followings:

- For part 1; Not applicable.
- For part 2; Accumulation ratios: Ro[AUC(0- $\tau$ )], R(Cmax), R(C $\tau$ ).

#### 9.2.3 Population of Interest

The secondary pharmacokinetic analyses will be based on the Pharmacokinetic population, unless otherwise specified.

### 9.2.4 Strategy for Intercurrent (Post-Randomization) Events

Not applicable.

# 9.2.5 Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 12: List of Data Displays and will be based on GSK Data Standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 9.2.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

#### **Statistical Methodology Specification**

#### **Part 2 Steady State Assessments**

#### **Endpoint / Variables**

GSK2838232 pre-dose values between Days 2 through 11

#### **Model Specification**

• Achievement of plasma GSK2838232 steady-state will be assessed by calculating the 90% CI of the slope of the linear regression of  $\log_e(C\tau)$  versus time. The dependent variable in the mixed effect model will be  $\log_e(C\tau)$  and the model will include a random intercept effect for participant and a fixed slope effect for study day. Day will be treated as a continuous variable in the model.

#### **Model Checking & Diagnostics**

- Model assumptions will be applied, but appropriate adjustments may be made based on the data.
- The Kenward and Roger method for approximating the denominator degrees of freedom and correcting for bias in the estimated variance-covariance of the fixed effects will be used.
- An unstructured covariance structure for the R matrix will be used by specifying 'type=UN' on the REPEATED line.
- In the event that this model fails to converge, alternative correlation structures may be considered such as CSH or CS.
- Akaike's Information Criteria (AIC) will be used to assist with the selection of covariance structure.
- Normality assumptions underlying the model used for analysis will be examined by obtaining a
  normal probability plot of the residuals and a plot of the residuals versus the fitted values (i.e.
  checking the normality assumption and constant variance assumption of the model
  respectively) to gain confidence that the model assumptions are reasonable.
- If there are any departures from the distributional assumptions, alternative models will be explored using appropriate transformed data.

#### Model Results Presentation

- Steady state will be reached if the pre-dose concentration slope estimate is close to zero or the 90% CI for the slope estimate includes zero.
- Mean plasma GSK2838232 pre-dose values between Days 2 through 11 and  $C_{\tau}$  of Day 11 will be plotted against time on linear and semi-logarithmic scale..

#### **Subgroup Analyses**

Not applicable

### **Sensitivity and Supportive Analyses**

Not applicable

#### Part 2 Accumulation

#### **Endpoint / Variables**

AUC(0-τ), Cmax and Cτ between Day 11 and Day 1

#### Model Specification

• The extent of accumulation of GSK2838232 will be evaluated by comparing AUC(0- $\tau$ ), Cmax and C $\tau$  between Day 11 and Day 1. For each of these comparisons an analysis of variance will be conducted on the log scale. The difference between Day 11 and Day 1 least square (LS) means and a 90% CI will be computed by fitting a mixed effects model with the log-transformed PK parameter as the dependent variable, day as a fixed effect and participant as a random effect.

#### **Model Checking & Diagnostics**

- Model assumptions will be applied, but appropriate adjustments may be made based on the data
- The Kenward and Roger method for approximating the denominator degrees of freedom and correcting for bias in the estimated variance-covariance of the fixed effects will be used.
- Normality assumptions underlying the model used for analysis will be examined by obtaining a
  normal probability plot of the residuals and a plot of the residuals versus the fitted values (i.e.
  checking the normality assumption and constant variance assumption of the model
  respectively) to gain confidence that the model assumptions are reasonable.
- If there are any departures from the distributional assumptions, alternative models will be explored using appropriate transformed data.

#### **Model Results Presentation**

- Geometric least-squares means for each treatment, point estimates and associated 90% confidence intervals for the ratios for each parameter will be produced in tabular format.
   Estimates of within-subject variability (%CVw) will also be provided. %CVw represents a pooled measure of within-subject variability across all treatments.
- Comparative plots of individual Accumulation Ratio will be generated by dose group on linear and semi-logarithmic scales.
- The accumulation ratio will be listed and summarized along with other PK parameters.
- Supportive SAS output from statistical analysis will be generated.

## **Subgroup Analyses**

Not applicable

## **Sensitivity and Supportive Analyses**

Not applicable

# 9.3 Exploratory Pharmacokinetic Analyses

Not applicable.

# 10. POPULATION PHARMACOKINETIC (POPPK) ANALYSES

Not applicable.

#### 11. PHARMACODYNAMIC ANALYSES

Not applicable.

# 12. PHARMACOKINETIC / PHARMACODYNAMIC ANALYSES

Not applicable.

#### 13. REFERENCES

GlaxoSmithKline documents:

GUI 51487: Non-compartmental Analysis of Pharmacokinetic Data, CPMS Global

Reporting and Analysis Plan (RAP) Template [Phases I to IV] Version 2.0 [Dated: 08-AUG-2017]

#### 14. APPENDICES

# 14.1 Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population

# 14.2.1 Exclusions from Per Protocol Population

Not applicable.

# 14.2 Appendix 2: Schedule of Activities

# 14.2.1 Protocol Defined Schedule of Events

## Schedule of Assessments for Part 1A and Part 1B: Single Dose RBA $\pm$ Food

| | Screening<br>(within 30 days of | in 30 days of | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | Day 1 - carried out<br>over multiple days –<br>except as noted in | Day -3 | Day -2 | Day -1 | Day 1 | Day 2 | Day 3 | Day 4 | Day 5 | Day 6 | Day 7 | 7-14<br>days |
| | footnotes) | | | | | 24 h | 48 h | 72 h | 96 h | 120 h | | |
| Admission to Unit | | X2 | | | | | | | | | | |
| Outpatient Visit | Χ | | | | | | | | | | | X |
| Informed Consent | Χ | | | | | | | | | | | |
| Medical/medication/ | | | | | | | | | | | | |
| drug/alcohol history | Χ | | | | | | | | | | | |
| (Demographics) | | | | | | | | | | | | |
| Full Physical Examination | Х | | | | | | | | | | | |
| Brief Physical Examination | | | Х | | | | X | | | | | X |
| Height, Weight, BMI | Χ | | | | | | | | | | | |
| Inclusion/Exclusion | Χ | | | | | | | | | | | |
| Vital signs <sup>3</sup> | Χ | | X | X | X | X | Χ | Χ | | | | X |
| 12 Lead ECG <sup>4</sup> | Χ | | Х | Χ | Х | Χ | Χ | | | | | Х |
| Echocardiogram <sup>5</sup> | Χ | | | | | | | | | | | |
| Drug/alcohol/cotinine screen | Χ | Χ | | | | | | | | | | |
| HbsAg, HCV, HIV tests | Χ | | | | | | | | | | | |
| Hem/Chem/Urine tests <sup>6</sup> | Χ | | Х | Х | | Х | | Х | | | | Х |
| Serum FSH (as appropriate) | Χ | | | | | | | | | | | |
| Troponin I <sup>7</sup> | Χ | | | X | Х | Χ | | X | | | | |
| 24 h Holter Monitoring <sup>8</sup> | Χ | | | | | | | | | | | |
| Pregnancy test (women) | Χ | Χ | | | | | | | | | | Χ |
| Run-in Dosing with RTV | | | Х | Х | | | | | | | | |
| Dosing with GSK2838232+RTV | | | | | X | | | | | | | |

| | Screening<br>(within 30 days of | Periods 1 | Periods 1 through 3 | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | Day 1 - carried out<br>over multiple days –<br>except as noted in | Day -3 | B Day -2 | Day -1 | Day 1 | Day 2 | Day 3 | Day 4 | Day 5 | Day 6 | Day 7 | 7-14<br>days |
| | footnotes) | | | | | 24 h | 48 h | 72 h | 96 h | 120 h | | |
| PK Sampling <sup>9</sup> | | | | | X | Χ | Х | Χ | Χ | Χ | | |
| Adverse Event Review <sup>10</sup> | | | | Х | Χ | Х | Х | Х | Х | Х | Х | Х |
| Con Med Review | | | Х | Х | Χ | Χ | Х | Χ | Χ | Χ | Χ | Χ |
| Discharge from Unit <sup>11</sup> | | | | | | Х | | | | | | |
| Out Patient Visit | | | | | | | Х | Χ | Х | Χ | Χ | |

205820

BMI = Body Mass Index; ECG = Electrocardiogram; FSH = Follicle Stimulating; HbsAg = Hepatitis B surface Antigen; HCV = Hepatitis C Virus; HIV = Human Immunodeficiency Virus; Hem/Chem = Hematology/Clinical Chemistry; RTV = Ritonavir; PK = Pharmacokinetic(s); Con Med = Concomitant medications.

- 1. Follow-up Visit to take place after Treatment Period 2.
- 2. When participants stay in the unit across treatment periods, drug/alcohol/cotinine screen and pregnancy test (women) are not required on Day -3 for later periods.
- 3. On Day 1, Blood pressure (BP) and Heart rate (HR) will be collected at pre-dose (triplicate) and single assessments at 1, 2, 4, 6, 8, 12, 24, 48, and 72 h post-dose.
- 4. On Day 1, 12-lead ECG will be collected at pre-dose (triplicate), and single assessments at 1, 2, 4, 6, 8, 12, 24, 48 and 72 h post-dose.
- 5. Echocardiograms must be within 100 days of Day 1.
- 6. Samples for Chemistry and Hematology: Blood samples will be obtained after an 8-hour fast.
- 7. Collect one troponin sample to be analyzed at local laboratory. A second sample will be collected, frozen and stored on site for potential high sensitivity troponin analysis.
- 8. 24-h Holter monitoring to be performed after confirming negative urine drug screen at screening, and must be within 30 days of Day 1. Holter monitoring on other days only if needed.
- 9. Plasma PK samples for bioanalysis for GSK2838232 will be collected pre-dose (within 15 minutes prior to dosing) and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, 36, 48, 72, 96, and 120 h post-dose. Samples will be acidified with an equal volume of 50 mmol citrate acid buffer pH 4.0.
- 10. An AE enquiry will be made at each visit, participants will be asked if they have experienced any neuropsychiatric adverse events, including psychosis or altered mental status. (see guidance for grading Altered Mental Status in Appendix 4).
- 11. Participants may be discharged after all study procedures are completed. Participants will be in house for PK blood samples on Day 3 (48 h), Day 4 (72 h), Day 5 (96 h) and Day 6 (120 h) of both study periods.

# Schedule of Assessments for Part 2: Repeated Doses for 11 days:

| Measurement | Screening<br>(within 30<br>days of Day<br>1 - carried<br>out over | | | | | | | | | | | | | | | | | | Follow-<br>up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Measurement | multiple days | Day<br>–1 | Day<br>1 | Day<br>2 | Day<br>3 | Day<br>4 | Day<br>5 | Day<br>6 | Day<br>7 | Day<br>8 | Day<br>9 | Day<br>10 | Day<br>11<br>0 h | Day<br>12<br>24 h | Day<br>13<br>48 h | Day<br>14<br>72 h | Day<br>15<br>96 h | Day<br>16<br>120<br>h | 7-14<br>days<br>after<br>last<br>dose |
| Admission to Unit | | Χ | | | | | | | | | | | | | | | | | |
| Informed Consent | X | | | | | | | | | | | | | | | | | | |
| Medical/medication/<br>drug/alcohol history<br>(Demographics) | X | | | | | | | | | | | | | | | | | | |
| Full Physical Examination | X | | | | | | | | | | | | | Х | | | | | |
| Brief Physical Examination | | Х | | | | | | | | | | | | | | | | | Х |
| Height, Weight, BMI | X | | | | | | | | | | | | | | | | | | |
| Inclusion/Exclusion | X | | | | | | | | | | | | | | | | | | |
| Medical History | Х | | | | | | | | | | | | | | | | | | |
| Vital Signs <sup>1</sup> | Х | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | | | Χ |
| 12-lead ECG <sup>2</sup> | X | Χ | Χ | Χ | Χ | | Х | | | Х | | | Х | X | | | | | Χ |
| Echocardiogram <sup>3</sup> | X | | | | | | | | | | | | | | | | | | |
| Drug/alcohol/ /cotinine<br>Screen | X | Х | | | | | | | | | | | | | | | | | |
| HbsAg, HCV, HIV<br>Testing | Х | | | | | | | | | | | | | | | | | | |
| Hem/Chem tests <sup>4</sup> | Х | Χ | | Χ | | Х | | Х | | Х | | | Χ | | | Х | | | Χ |
| Urinalysis | Х | Χ | | Χ | | Χ | | | | | | | Х | | | Х | | | Χ |
| Serum FSH (as appropriate) | Х | | | | | | | | | | | | | | | | | | |
| Troponin I <sup>5</sup> | Х | Χ | Χ | Χ | | | Х | | | Х | | | Х | | | Х | | | |

| | Screening<br>(within 30<br>days of Day<br>1 - carried | | | | | | | | | | | | | | | | | | Follow-<br>up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Measurement | out over<br>multiple days<br>- except as<br>noted in<br>footnotes) | Day<br>-1 | Day<br>1 | Day<br>2 | Day<br>3 | Day<br>4 | Day<br>5 | Day<br>6 | Day<br>7 | Day<br>8 | Day<br>9 | Day<br>10 | Day<br>11<br>0 h | Day<br>12<br>24 h | Day<br>13<br>48 h | Day<br>14<br>72 h | Day<br>15<br>96 h | Day<br>16<br>120<br>h | 7-14<br>days<br>after<br>last<br>dose |
| 24 h Holter Monitoring <sup>6</sup> | Х | | | | | | | | | | | | | | | | | | |
| Pregnancy Test (females) | Х | Х | | | | | | | | | | | | | | | | | Х |
| Dosing of GSK2838232 | | | Χ | Χ | Х | Χ | Х | Х | Χ | Χ | Χ | Χ | Х | | | | | | |
| Plasma PK sampling <sup>7</sup> | | | Х | Χ | Χ | Χ | Х | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Х | Χ | Х | Χ | |
| Adverse Event<br>Assessment <sup>8</sup> | | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| Concomitant<br>Medications | | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| Discharge from Unit | | | | | | | | | | | | | | | X <sup>9</sup> | | | | |
| Out Patient Visit | Х | | | | | | | | | | | | | | | Χ | Χ | Χ | Х |

BMI = Body Mass Index; ECG = Electrocardiogram; FSH = Follicle Stimulating Hormone; HbsAg = Hepatitis B surface Antigen; HCV = Hepatitis C Virus; Hem/Chem = Hematology/Clinical Chemistry; HIV = Human Immunodeficiency Virus; IP = Investigational Product; PK = Pharmacokinetic(s).

- 1. A single blood pressure (BP) and Heart rate (HR) assessment will be collected at screening and Day -1. On Day 1 triplicate BP and HR will be collected at pre-dose and single assessments at 1, 4, 24, 48 and 72 h (Day 4) post-dose, Day 5, Day 6, Day 7, Day 8, Day 9, Day 10, Day 11 at pre-dose (triplicate), and single assessment at 1, 4, 24, 48 and 72 h post-dose, and at follow-up.
- 2. A single 12-Lead ECG will be collected at screening and Day -1. On Day 1 triplicate 12-Lead ECGs will be collected at pre-dose, and then single 12-Lead ECGs at 1, 4 and 12 h post-dose. Single 12-Lead ECGs will be collected on Days 2, 3, 5, 8. On Day 11 triplicate 12-Lead ECGs will be collected pre-dose, and then single 12-Lead ECGs collected at 1, 4, 12 and 24 h post-dose and at follow-up.
- 3. Echocardiograms must be within 100 days of Day 1.
- 4. Samples for Chemistry and Hematology: Blood samples will be obtained after an 8-hour fast.
- 5. Collect one troponin sample to be analyzed at local laboratory. A second sample will be collected and frozen for potential high sensitivity troponin analysis.
- 6. 24-h Holter monitoring to be performed after confirming negative urine drug screen at screening, and must be within 30 days of Day 1. Holter monitoring on other days only if needed.

- 7. Plasma PK samples for GSK2838232 will be collected as follows: Day 1; pre-dose (within 15 minutes prior to dosing) and 0.5,1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12 and 24 h post-dose (prior to Day 2 dose). Days 3 to 10 pre-dose (within 15 minutes prior to dosing). Day 11; pre-dose (within 15 minutes prior to dosing) and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, 36, 48, 72, 96 and 120 h post-dose. Samples will be acidified with an equal volume of 50 mmol citrate acid buffer pH 4.0.
- 8. An AE enquiry will be made at each visit, participants will be asked if they have experienced any neuropsychiatric adverse events, including psychosis or altered mental status. (see guidance for grading Altered Mental Status in Appendix 4).
- 9. Participants will be discharged after all study procedures are completed on the morning of Day 13 (after the 48 h post-final dose sample time point) with instructions to return fasted on the mornings of Day 14 for 72 h PK sample, Day 15 for 96 h PK sample, and Day 16 for 120 h PK sample

2017N322544\_01 **CONFIDENTIAL** 

# 14.3 Appendix 3: Assessment Windows

# 14.3.1 Definitions of Assessment Windows for Analyses

Not applicable.

2017N322544\_01 **CONFIDENTIAL** 

# 14.4 Appendix 4: Study Phases and Treatment Emergent Adverse Events

## 14.4.1 Study Phases

Assessments and events will be classified according to the time of occurrence relative to study treatment.

| Treatment Phase | Definition |
|---|---|
| Pre-Treatment | Date/Time < Study Treatment Start Date/Time |
| On- Treatment | Study Treatment Start Date/Time ≤ Date/Time ≤ Study Treatment Stop Date/Time |
| Post- Treatment | Date/Time > Study Treatment Stop Date/Time |

### 14.4.4.1 Study Phases for Concomitant Medication

| Study Phase | Definition |
|---|---|
| Prior | If medication end date is not missing and is before 28 days prior to screening visit |
| Concomitant | Any medication that is not a prior |

#### NOTES:

 Please refer to Appendix 7: Reporting Standards for Missing Data for handling of missing and partial dates for concomitant medication. Use the rules in this table if concomitant medication date is completely missing.

# 14.4.2 Treatment Emergent Flag for Adverse Events

| Flag | Definition |
|---|---|
| Treatment<br>Emergent | If AE onset date is on or after treatment start date & on or before treatment stop date. (plus washout or protocol-specified time limit (e.g. half-life of drug, certain number of days, etc.). |
| | Study Treatment Start Date/Time ≤ AE Start Date/Time. |
| | <ul> <li>For studies with greater than one treatment period (e.g., crossover study), if AE onset is during one period and worsens during a later period it would be counted in both periods. For the initial period the logic would be as above. For the later period the logic would use the treatment dates associated with the later period:</li> </ul> |
| | <ul> <li>Treatment Period Start Date ≤ AE Worsening Date.</li> </ul> |

#### NOTES:

- If the study treatment stop date is missing, then the AE will be considered to be On-Treatment.
- Time of study treatment dosing and start/stop time of AEs should be considered, if collected.

# 14.4.3 Adverse Events Assignment to Treatment Period for Part 1

Adverse events (AEs) will be assigned to a treatment period and corresponding treatment received in that treatment period after the imputations defined in RAP section 14.7.3 have been performed.

35

- Treatment Period 1: all AEs with start date/time at the time of or after IMP administration in Treatment Period 1 and before IMP administration in Treatment Period 2
- Treatment Period 2: all AEs with start date/time at the time of or after IMP administration in Treatment Period 2 and before IMP administration in Treatment Period 3
- Treatment Period 3: all AEs with start date/time at the time of or after IMP administration in Treatment Period 3

Thus, AEs occurring during the 1<sup>st</sup> washout will be assigned to the treatment received in Treatment Period 1, AEs occurring during the 2<sup>th</sup> washout will be assigned to the treatment received in Treatment Period 2 and AEs occurring during follow-up will be assigned to the treatment received in Treatment Period 3.

# 14.4.4 Concomitant Medication Assignment to Treatment Period for Part 1

Concomitant medications (CMs) will be assigned to a treatment period and corresponding treatment received in that treatment period after the imputations defined in RAP section 14.7.3 have been performed.

- Treatment Period 1: all CMs with start date/time at the time of or after IMP administration in Treatment Period 1 and before IMP administration in Treatment Period 2
- Treatment Period 2: all CMs with start date/time at the time of or after IMP administration in Treatment Period 2 and before IMP administration in Treatment Period 3
- Treatment Period 3: all CMs with start date/time at the time of or after IMP administration in Treatment Period 3

Thus, CMs occurring during the 1<sup>st</sup> washout will be assigned to the treatment received in Treatment Period 1, CMs occurring during the 2<sup>th</sup> washout will be assigned to the treatment received in Treatment Period 2 and CMs occurring during follow-up will be assigned to the treatment received in Treatment Period 3.

36
# 14.5 Appendix 5: Data Display Standards & Handling Conventions

### 14.5.1 Reporting Process

#### Software

The currently supported versions of SAS and WinNonlin software will be used.

#### **Analysis Datasets**

- Analysis datasets will be created according to AdaM IG Version 1.1.
- For creation of ADaM datasets (ADCM/ADAE), the same version of dictionary datasets will be implemented for conversion from SI to SDTM.
- Define XML Version 2.0

#### **Generation of RTF Files**

RTF files will be generated for Tables, Listings, and Figures, one RTF file per item.

### 14.5.2 Reporting Standards

#### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated:
  - 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings
  - 6.01 to 6.11: Principles Related to Summary Tables
  - 7.01 to 7.13: Principles Related to Graphics
- Do not include participant level listings in the main body of the GSK Clinical Study Report. All
  participant level listings should be located in the modular appendices as ICH or non-ICH
  listings

#### **Formats**

- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of decimal places (DP's).

#### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses:
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the participant's listings.

#### **Unscheduled Visits**

| Unscheduled visits will not be included in summary tables and/or figures. | |
|---|---|
| All unscheduled visits will be included in listings. | |
| Descriptive Summar | Descriptive Summary Statistics |
| Continuous Data | Refer to IDSL Statistical Principle 6.06.1 |
| Categorical Data N, n, frequency, % | |
| Graphical Displays | |

- Refer to IDSL Statistical Principals 7.01 to 7.13
- The same symbol and line type will be used across figures to represent a given treatment group. The placebo group will be displayed using symbol type=empty circle and line type= solid line and color=black.
- When line plots are presented with treatment groups overlaid, the x-values will be offset (jittered) so the data are not plotted on top of each other.
- X-axis variables of time and dose will be plotted as continuous numeric variables...

### 14.5.3 Reporting Standards for Pharmacokinetic Data

| Pharmacokinetic Concentration Data | |
|---|---|
| PC Windows Non-<br>Linear (WNL) File | PC WNL file (CSV format) for the non compartmental analysis by Clinical Pharmacology Modelling and Simulation function will be created according to Standards for the Transfer and Reporting of PK Data using HARP. Note: Concentration values will be imputed as per GUI_51487 |
| Descriptive Summary<br>Statistics, Graphical<br>Displays and Listings | Refer to IDSL PK Display Standards. Refer to IDSL Statistical Principle 6.06.1. Note: Concentration values will be imputed as per GUI_51487 for descriptive summary statistics/analysis and summarized graphical displays only. |
| Pharmacokinetic Para | ameter Derivation |
| PK Parameter to be<br>Derived by<br>Programmer | The following PK parameters will be derived by the Programmer: C24, C $\tau$ , Ctrough. Ro[AUC(0- $\tau$ )], R(Cmax), R(C $\tau$ ) |
| Pharmacokinetic Para | Pharmacokinetic Parameter Data |
| Is NQ impacted PK<br>Parameters Rule<br>Being Followed | No |
| Descriptive Summary<br>Statistics, Graphical<br>Displays and Listings | Refer to IDSL PK Display Standards. |

| Descriptive Summary Statistics | |
|---|---|
| Continuous Data | Refer to IDSL Statistical Principle 6.06.1 |
| Categorical Data | N, n, frequency, % |
| Reporting of Pharmacokinetic Concentration Data | |
| Descriptive Summary | Refer to IDSL Statistical Principle 6.06.1 |
| Statistics | Assign zero to NQ values (Refer to GUI_51487 for further details) |

| Reporting of Pharmaco | Reporting of Pharmacokinetic Parameters |
|---|---|
| Descriptive Summary<br>Statistics (Loge<br>Transformed) | <ul> <li>N, n, geometric mean, 95% CI of geometric mean, standard deviation (SD) of logged data and between and or within geometric coefficient of variation (CVb/w (%)) will be reported.</li> <li>[1] Geometric mean = exp(mean log<sub>e</sub>-transformed values)</li> <li>[2] CV<sub>b</sub> (%) = √ (exp(SD²) - 1) * 100 (SD = SD of log transformed data)</li> <li>[3] CV<sub>w</sub> (%) = √ (exp(MSE) - 1) * 100 (MSE = mean square error from mixed effect model of loge-transformed data).</li> </ul> |
| All Parameters | N, n, mean, SD, median, minimum, maximum |
| Summary Tables | The following PK parameters will not be summarised: %AUCex |
| Listings | Additionally, include the first point, last point and number of points used in the determination of lambda_z for listings. |

### **Graphical Displays**

- Refer to IDSL Statistical Principals 7.01 to 7.13.
- The same symbol and line type will be used across figures to represent a given treatment group. The placebo group will be displayed using symbol type=empty circle and line type= solid line and color=black.
- When line plots are presented with treatment groups overlaid, the x-values will be offset (jittered) so the data are not plotted on top of each other.
- X-axis variables of time and dose will be plotted as continuous numeric variables.

#### 14.6 Appendix 6: Derived and Transformed Data

#### 14.6.1 General

#### **Multiple Measurements at One Time Point**

- Mean of the measurements will be calculated and used in any derivation of summary statistics but if listed, all data will be presented.
- If there are two values within a time window (as per Section 14.3.1) the value closest to the target day for that window will be used. If values are the same distance from the target, then the mean will be taken.
- Participants having both High and Low values for Normal Ranges at any post-baseline visits for safety parameters will be counted in both the High and Low categories of "Any visit post-baseline" row of related summary tables. This will also be applicable to relevant Potential Clinical Importance summary tables.

#### Study Day

- Calculated as the number of days from First Dose Date:
  - Ref Date = Missing → Study Day = Missing
  - Ref Date < First Dose Date → Study Day = Ref Date First Dose Date</li>
  - Ref Data ≥ First Dose Date → Study Day = Ref Date (First Dose Date) + 1

### 14.6.2 Study Population

#### **Demographics**

#### Age

- GSK standard IDSL algorithms will be used for calculating age where birth date will be imputed as follows:
  - Any participant with a missing day will have this imputed as day '15'.
  - Any participant with a missing date and month will have this imputed as '30th June'.
  - The age will be calculated by Data Management and mapped from ClinBase to SDTM dataset DM
- Birth date will be presented in listings as 'YYYY'.

#### **Body Mass Index (BMI)**

Calculated as Weight (kg) / [Height (m)]<sup>2</sup>

#### **Treatment Compliance**

Treatment compliance will be calculated based on the formula:

## Treatment Compliance = Number of Actual Doses / (Planned Treatment Duration in Days \* Frequency)

- Frequency is 2 for BID and 1 for QD. Treatment compliance could be greater than 100% if there are events of overdose. Cumulative compliance (since Day 1) at each visit will be calculated.
- Planned Treatment Duration is defined as 1 day for study part 1, and as 11 day for study part 2.

#### **Extent of Exposure**

- Number of days of exposure to study drug will be calculated based on the formula:
   Duration of Exposure in Days = Treatment Stop Date (Treatment Start Date) + 1
- Participants who were randomized but did not report a treatment start date will be categorised

#### **Demographics**

as having zero days of exposure.

• The cumulative dose will be based on the formula:

**Cumulative Dose = Sum of (Number of Days x Total Daily Dose)** 

• If there are any treatment breaks during the study, exposure data will be adjusted accordingly.

### 14.6.3 Efficacy

Not applicable.

### 14.6.4 Safety

#### **ECG Parameters**

#### **RR** Interval

- IF RR interval (msec) is not provided directly, then RR can be derived as :
  - [1] If QTcB is machine read & QTcF is not provided, then:

$$RR = \left[ \left( \frac{QT}{QTcB} \right)^2 \right] * 1000$$

[2] If QTcF is machine read and QTcB is not provided, then:

$$RR = \left[ \left( \frac{QT}{QTcF} \right)^3 \right] * 1000$$

 If ECGs are manually read, the RR value preceding the measurement QT interval should be a collected value THEN do not derive.

#### **Corrected QT Intervals**

- When not entered directly in the eCRF, corrected QT intervals by Bazett's (QTcB) and Fredericia's (QTcF) formulas will be calculated, in msec, depending on the availability of other measurements.
- IF RR interval (msec) is provided then missing QTcB and/or QTcF will be derived as :

$$QTcB = \frac{QT}{\sqrt{\frac{RR}{1000}}}$$

$$QTcF = \frac{QT}{3\sqrt{\frac{RR}{1000}}}$$

Also QTc interval will be categorized as follows:

| ECG Parameter | Potential Clinical Importance Range (PCI) | Units |
|---|---|---|
| LOO I didilictei | 1 otential official importance range (1 of) | Office |
| Absolute QTc Interval | >450 to ≤480 | msec |
| Absolute QTc Interval | >480 to ≤500 | msec |
| Absolute QTc Interval | >500 | msec |
| Increase from Baseline QTc | ≤30 | msec |
| Increase from Baseline QTc | >30 to ≤60 | msec |
| Increase from Baseline QTc | >60 | msec |

#### **Laboratory Parameters**

• If a laboratory value which is expected to have a numeric value for summary purposes, has a non-detectable level reported in the database, where the numeric value is missing, but typically a character value starting with '<x' or '>x' (or indicated as less than x or greater than x in the comment field) is present, will be imputed with the value of the number without the sign for the descriptive statistics and the calculation of changes from baseline, e.g., a value of <2.2 will be imputed as 2.2 for the calculations. There will be no imputation in the data listings; all values will be displayed as recorded in the database.

#### 14.6.5 Pharmacokinetic

Calculation of Pharmacokinetic Parameter Values Not Described in Section 9 (refer to GUI\_51487 for pharmacokinetic analysis information)

#### lambda\_z (terminal phase rate constant)

 Slope of the line determined by linear regression of logarithmically transformed concentration v. time data

#### %AUCex (percentage of AUC(0-∞) obtained by extrapolation)

Calculated as 100 x [AUC(0-∞) – AUC(0-t)] / AUC(0-∞)

### 14.6.6 Population Pharmacokinetic (PopPK)

Not applicable.

### 14.6.7 Pharmacodynamic

Not applicable.

### 14.7 Appendix 7: Reporting Standards for Missing Data

### 14.7.1 Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | Participant study completion (i.e. as specified in the protocol) was defined as participants who has received the study treatment per the protocol and who has completed all phases of the study including the follow-up visit. The study including the follow-up visit. |
| | The end of the study is defined as the last participant's last visit. |
| | Withdrawn participants will not be replaced in the study. |
| | All available data from participants who were withdrawn from the study will be listed and all available planned data will be included in summary tables and figures, unless otherwise specified. |
| | Withdrawal visits will be summarised as withdrawal visits. |

### 14.7.2 Handling of Missing Data

| Reporting Detail |
|---|
| <ul> <li>Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument:</li> <li>These data will be indicated by the use of a "blank" in participant listing displays. Unless all data for a specific visit are missing in which case the data is excluded from the table.</li> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to be missing data and should be displayed as such.</li> </ul> |
| Any participants excluded from the summaries and/or statistical analyses will be documented along with the reason for exclusion in the clinical study report. |

### 14.7.3 Handling of Missing and Partial Dates

| Element | Reporting Detail |
|---|---|
| General | Partial dates will be displayed as captured in participant listing displays. |
| Adverse<br>Events | <ul> <li>The eCRF allows for the possibility of partial dates (i.e., only month and year) to be recorded for AE start and end dates; that is, the day of the month may be missing. In such a case, the following conventions will be applied for calculating the time to onset and the duration of the event: <ul> <li>Missing Start Day: First of the month will be used unless this is before the start date of study treatment; in this case the study treatment start date will be used and hence the event is considered On-treatment as per Appendix: Treatment States and Phases.</li> <li>Missing Stop Day: Last day of the month will be used, unless this is after the stop date of study treatment; in this case the study treatment stop date will be used.</li> </ul> </li> <li>Completely missing start or end dates (i.e. no year specified) will remain</li> </ul> |

| Element | Reporting Detail |
|---|---|
| | missing, with no imputation applied. Consequently, time to onset and duration of such events will be missing. |
| Element | Reporting Detail |
| Concomitant<br>Medications/<br>Medical<br>History | <ul> <li>imputed using the following convention:</li> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month</li> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month.</li> </ul> |
| | The recorded partial date will be displayed in listings. |

### 14.8 Appendix 8: Values of Potential Clinical Importance

### 14.8.1 Laboratory Values

Division of AIDS (DAIDS, Version 2.0, November 2014) AE grades 2, 3, and 4 of lab abnormalities will be listed by subject, period/treatment, visit, and actual date and time.

| Haematology | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| | | Male | | 0.54 |
| Hematocrit | Ratio of 1 | Female | | 0.54 |
| | | $\Delta$ from BL | ↓0.075 | |
| | - // | Male | | 180 |
| Hemoglobin | g/L | Female | | 180 |
| | | $\Delta$ from BL | <b>↓25</b> | |
| Lymphocytes | x10 <sup>9</sup> / L | | 0.8 | |
| Neutrophil Count | x109/ L | | 1.5 | |
| Platelet Count | x109/ L | | 100 | 550 |
| While Blood Cell Count (WBC) | x10 <sup>9</sup> / L | | 3 | 20 |

| Clinical Chemistry | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| Albumin | g/L | | 30 | |
| Calcium | mmol/L | | 2 | 2.75 |
| Creatinine | $\mu$ mol/L | $\Delta$ from BL | | <b>↑ 44.2</b> |
| Glucose | mmol/L | | 3 | 9 |
| Magnesium | mmol/L | | 0.5 | 1.23 |
| Phosphorus | mmol/L | | 0.8 | 1.6 |
| Potassium | mmol/L | | 3 | 5.5 |
| Sodium | mmol/L | | 130 | 150 |
| Total CO2 | mmol/L | | 18 | 32 |

| Liver Function | | | |
|---|---|---|---|
| Test Analyte | Units | Category | Potential Clinical Importance Range |
| ALT/SGPT | U/L | High | ≥ 2x ULN |
| AST/SGOT | U/L | High | ≥ 2x ULN |
| AlkPhos | U/L | High | ≥ 2x ULN |
| T Bilirubin | µmol/L | High | ≥ 1.5xULN |
| | µmol/L | | 1.5xULN T. Bilirubin |
| T. Bilirubin + ALT | | High | + |
| | U/L | | ≥ 2x ULN ALT |

### 14.8.2 ECG

| ECG Parameter | Units | Potential Clinical Importance Range | |
|---|---|---|---|
| | | Lower | Upper |
| Absolute | Absolute | | |
| Absolute QTc Interval | msec | | > 450 |
| Absolute PR Interval | msec | < 110 | > 220 |
| Absolute QRS Interval | msec | < 75 | > 110 |
| Change from Baseline | | | |
| Increase from Baseline QTc | msec | | > 60 |

### 14.8.3 Vital Signs

| Vital Sign Parameter Units | | Potential Clinical Importance Range | |
|---|---|---|---|
| (Absolute) | | Lower ( <x)< th=""><th>Upper (&gt;x)</th></x)<> | Upper (>x) |
| Systolic Blood Pressure | mmHg | < 85 | > 160 |
| Diastolic Blood Pressure | mmHg | < 45 | > 100 |
| Heart Rate | bpm | < 40 | > 110 |

14.9 Appendix 9: Population Pharmacokinetic (PopPK) Analyses

- **14.9.1** Population Pharmacokinetic (PopPK) Dataset Specification Not applicable.
- **14.9.2** Population Pharmacokinetic (PopPK) Methodology Not applicable.

# 14.10 Appendix 10: Pharmacokinetic / Pharmacodynamic Analyses

- **14.10.1** Pharmacokinetic / Pharmacodynamic Dataset Specification Not applicable.
- **14.10.2** Pharmacokinetic / Pharmacodynamic Methodology Not applicable.

### 14.11 Appendix 11: Abbreviations & Trade Marks

### 14.11.1 Abbreviations

| Abbreviation | Description |
|---|---|
| A&R | Analysis and Reporting |
| ADaM | Analysis Data Model |
| AE | Adverse Event |
| AlkPhos | Alkaline Phosphatase |
| ALT | Alanine Aminotransferase |
| ANOVA | Analysis of Variance |
| AST | Aspartate Aminotransferase |
| ATC | Anatomical, Therapeutical, Chemical |
| AUC | Area-under-the-curve |
| AUC(0-∞) | Area under the concentration-time curve extrapolated to infinity |
| AUC(0-last) | Area under the concentration-time curve from time zero to the time of the last |
| | quantifiable concentration |
| AUC(0-t) | Partial area under the concentration-time curve to time |
| BMI | Body Mass Index |
| BP | Blood Pressure |
| C24 | Observed concentration 24 hours post-dose, determined directly from the |
| | concentration-time data. |
| CDISC | Clinical Data Interchange Standards Consortium |
| Chem | Chemistry |
| CI | Confidence Interval |
| CL | Clearance |
| CM | Concomitant Medication |
| C <sub>max</sub> | Maximum observed concentration, determined directly from the concentration- |
| | time data. |
| CPMS | Clinical Pharmacology Modelling & Simulation |
| CS | Clinical Statistics |
| CSP | Clinical Study Protocol |
| CSR | Clinical Study Report |
| Сτ | Observed concentration at time τ |
| DLT | Dose-limiting Toxicity |
| DP | Decimal Places |
| ECG | Electrocardiogram |
| eCRF | Electronic Case Record Form |
| FDA | Food and Drug Administration |
| FSH | Follicle Stimulating Hormone |
| GSK | GlaxoSmithKline |
| GUI | Guidance |
| HBsAG | Hepatitis-B-Virus Surface Antigen |
| HCV | Hepatitis C virus |
| Hem | Hematology |
| HIV | Human Immunodeficiency Virus |

| Abbreviation | Description |
|---|---|
| IA | Interim Analysis |
| ICH | International Conference on Harmonisation |
| IDSL | Integrated Data Standards Library |
| IP | Investigational Product |
| Lambda_z | Terminal Phase Rate Constant |
| LOQ | Limit of Quantification |
| LS | Least Squares |
| MedDRA | Medical dictionary for Regulatory Activities |
| PCI | Potential Clinical Importance |
| PD | Pharmacodynamic |
| PDMP | Protocol Deviation Management Plan |
| PI | Principal Investigator |
| PK | Pharmacokinetics |
| PopPK | Population Pharmacokinetic |
| PP | Per Protocol |
| PT | Preferred Term |
| QCD | Quantitative Clinical Development |
| QD | Once daily |
| QTcB | Bazett's QT Interval Corrected for Heart Rate |
| QTcF | Frederica's QT Interval Corrected for Heart Rate |
| RAP | Reporting & Analysis Plan |
| Ro | Accumulation ratio |
| RTV | Ritonavir |
| SAC | Statistical Analysis Complete |
| SAE | Serious Adverse Event |
| SD | Standard deviation |
| SDTM | Study Data Tabulation Model |
| SGOT | Serum GlutamicOxaloacetic Transaminas |
| SGPT | Serum Glutamic-Pyruvic Transaminase |
| SOC | System Organ Class |
| SOP | Standard Operation Procedure |
| SRT | Safety Review Team |
| t <sub>1/2</sub> | Apparent terminal half-life |
| TA | Therapeutic Area |
| TFL | Tables, Figures & Listings |
| tlag | Lag-time (time delay between drug administration and first observed) |
| tlast | Time of last quantifiable concentration, determined directly from the |
| | concentration-time data. |
| tmax | Time to reach Cmax, determined directly from the concentration-time data. |

### 14.11.2 Trademarks

| Trademarks of the GlaxoSmithKline<br>Group of Companies |
|---------------------------------------------------------|
| Not applicable |

| Trademarks not owned by the GlaxoSmithKline Group of Companies |
|----------------------------------------------------------------|
| WinNonlin |
| SAS |
| Phoenix |

### 14.12 Appendix 12: List of Data Displays

### 14.12.1 Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|------------------|-------------------------|----------------|
| Study Population | 1.1 to 1.24 | Not applicable |
| Efficacy | Not applicable | Not applicable |
| Safety | 3.1 to 3.46 3.1 to 3.6 | |
| Pharmacokinetic | 5.1 to 5.18 5.1 to 5.23 | |
| Section | Listi | ings |
| ICH Listings | 1 to 67 | |
| Other Listings | 68 to 74 | |

### 14.12.2 Mock Example Shell Referencing

Non IDSL specifications will be referenced as indicated and if required an example mock-up displays provided in Appendix 13: Example Mock Shells for Data Displays.

| Section | Figure | Table | Listing |
|------------------|---------|---------|---------|
| Study Population | POP_Fn | POP_Tn | POP_Ln |
| Efficacy | EFF_Fn | EFF_Tn | EFF_Ln |
| Safety | SAFE_Fn | SAFE_Tn | SAFE_Ln |
| Pharmacokinetic | PK_Fn | PK_Tn | PK_Ln |

#### NOTES:

### 14.12.3 Deliverable [Priority]

| Delivery [Priority] [1] | Description |
|-------------------------|-------------------------------------|
| SAC [1] | Final Statistical Analysis Complete |

#### NOTES:

Non-Standard displays are indicated in the 'IDSL / Example Shell' or 'Programming Notes' column as '[Non-Standard] + Reference.'

<sup>1.</sup> Indicates priority (i.e. order) in which displays will be generated for the reporting effort.

### 14.12.4 Study Population Tables

| Study I | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Particip | ant Disposition | n | | | |
| 1.1. | Safety | ES8 | Summary of Participant Status and Reason for Study<br>Withdrawal – Part 1 | ICH E3, FDAAA, EudraCT Summarize by treatment /sequence and overall of each part | SAC [1] |
| 1.2. | Safety | ES8 | Summary of Participant Status and Reason for Study<br>Withdrawal – Part 2 | ICH E3, FDAAA, EudraCT Summarize by treatment /sequence and overall of each part | SAC [1] |
| 1.3. | Safety | SD1 | Summary of Treatment Status and Reasons for Discontinuation of Study Treatment – Part 1 | ICH E3 Summarize by treatment /sequence and overall of each part | SAC [1] |
| 1.4. | Safety | SD1 | Summary of Treatment Status and Reasons for Discontinuation of Study Treatment – Part 2 | ICH E3 Summarize by treatment /sequence and overall of each part | SAC [1] |
| 1.5. | Safety | ES4 | Summary of Participant Disposition at Each Study Epoch – Part 1 | ICH E3 | SAC [1] |
| 1.6. | Safety | ES4 | Summary of Participant Disposition at Each Study Epoch – Part 2 | ICH E3 | SAC [1] |
| 1.7. | Screened | ES6 | Summary of Screening Status and Reasons for Screen Failure – Part 1 | Journal Requirements | SAC [1] |
| 1.8. | Screened | ES6 | Summary of Screening Status and Reasons for Screen Failure – Part 2 | Journal Requirements | SAC [1] |

| Study F | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Protoco | ol Deviation | | | | |
| 1.9. | Safety | DV1 | Summary of Protocol Deviations – Part 1 | ICH E3 | SAC [1] |
| 1.10. | Safety | DV1 | Summary of Protocol Deviations – Part 2 | ICH E3 | SAC [1] |
| Popula | tion Analysed | | | | |
| 1.11. | Screened | SP1 | Summary of Study Populations – Part 1 | By treatment and combined overall | SAC [1] |
| 1.12. | Screened | SP1 | Summary of Study Populations – Part 2 | By treatment and combined overall | SAC [1] |
| Demog | raphic and Bas | eline Characteris | tics | | |
| 1.13. | Safety | DM3 | Summary of Demographic Characteristics – Part 1 | ICH E3, FDAAA, EudraCT | SAC [1] |
| 1.14. | Safety | DM1 | Summary of Demographic Characteristics – Part 2 | ICH E3, FDAAA, EudraCT | SAC [1] |
| 1.15. | Safety | DM11 | Summary of Age Ranges – Part 1 | EudraCT | SAC [1] |
| 1.16. | Safety | DM11 | Summary of Age Ranges – Part 2 | EudraCT | SAC [1] |
| 1.17. | Safety | DM5 | Summary of Race and Racial Combinations – Part 1 | ICH E3, FDA, FDAAA, EudraCT | SAC [1] |
| 1.18. | Safety | DM5 | Summary of Race and Racial Combinations – Part 2 | ICH E3, FDA, FDAAA, EudraCT | SAC [1] |
| Prior ar | Prior and Concomitant Medications | | | | |

| Study F | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 1.19. | Safety | MH4 | Summary of Medical Conditions – Part 1 | ICH E3. | SAC [1] |
| 1.20. | Safety | MH4 | Summary of Medical Conditions – Part 2 | ICH E3 | SAC [1] |
| 1.21. | Safety | CM1 | Summary of Concomitant Medications – Part 1 | ICH E3. | SAC [1] |
| 1.22. | Safety | CM1 | Summary of Concomitant Medications – Part 2 | ICH E3 | SAC [1] |
| Exposu | Exposure and Treatment Compliance | | | | |
| 1.23. | Safety | EX1 | Summary of Exposure to Study Treatment – Part 1 | ICH E3 | SAC [1] |
| 1.24. | Safety | EX1 | Summary of Exposure to Study Treatment – Part 2 | ICH E3 | SAC [1] |


205820

### 14.12.5 Efficacy Tables

Not applicable.

### 14.12.6 Efficacy Figures

Not applicable.

### 14.12.7 Safety Tables

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Advers | e Events (AEs) | | | | |
| 3.1. | Safety | AE5A | Summary of All Adverse Events by Maximum Intensity by System Organ Class and Preferred Term – Part 1 | ICH E3 Use AE5A/B (with a Total column across all grades/severities.) | SAC [1] |
| 3.2. | Safety | AE5A | Summary of All Adverse Events by Maximum Intensity by System Organ Class and Preferred Term – Part 2 | ICH E3 Use AE5A/B (with a Total column across all grades/severities.) | SAC [1] |
| 3.3. | Safety | AE3 | Summary of Common (>=5%) Adverse Events by Overall Frequency – Part 1 | ICH E3 | SAC [1] |
| 3.4. | Safety | AE3 | Summary of Common (>=5%) Adverse Events by Overall Frequency – Part 2 | ICH E3 | SAC [1] |
| 3.5. | Safety | AE5A | Summary of All Drug-Related Adverse Events by System Organ Class and Preferred Term and Maximum Intensity – Part 1 | ICH E3 | SAC [1] |
| 3.6. | Safety | AE5A | Summary of All Drug-Related Adverse Events by System Organ Class and Preferred Term and Maximum Intensity – Part 2 | ICH E3 | SAC [1] |
| 3.7. | Safety | AE15 | Summary of Common (>=5%) Non-serious Adverse Events by System Organ Class and Preferred Term (Number of Participant and Occurrences) – Part 1 | FDAAA, EudraCT | SAC [1] |
| 3.8. | Safety | AE15 | Summary of Common (>=5%) Non-serious Adverse Events by System Organ Class and Preferred Term (Number of Participant and Occurrences) – Part 2 | FDAAA, EudraCT | SAC [1] |

| Safety: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.9. | Safety | AE3 | Summary of Common (>=5%) Grade 2-4 Adverse Events by Overall Frequency – Part 1 | ICH E3 | SAC [1] |
| 3.10. | Safety | AE3 | Summary of Common (>=5%) Grade 2-4 Adverse Events by Overall Frequency – Part 2 | ICH E3 | SAC [1] |
| 3.11. | Safety | AE3 | Summary of Common (>=5%) Drug-Related Grade 2-4 Adverse Events by Overall Frequency – Part 1 | ICH E3 | SAC [1] |
| 3.12. | Safety | AE3 | Summary of Common (>=5%) Drug-Related Grade 2-4 Adverse Events by Overall Frequency – Part 2 | ICH E3 | SAC [1] |
| Serious | and Other Sig | nificant Adverse I | Events | | |
| 3.13. | Safety | AE16 | Summary of Serious Adverse Events by System Organ Class and Preferred Term (Number of Participants and Occurrences) – Part 1 | FDAAA, EudraCT | SAC [1] |
| 3.14. | Safety | AE16 | Summary of Serious Adverse Events by System Organ Class and Preferred Term (Number of Participants and Occurrences) – Part 2 | FDAAA, EudraCT | SAC [1] |
| 3.15. | Safety | AE1 | Summary of Adverse Events Leading to Permanent Discontinuation of Study Treatment or Withdrawal from Study by System Organ Class and Preferred Term /by Overall Frequency – Part 1 | IDSL | SAC [1] |
| 3.16. | Safety | AE1 | Summary of Adverse Events Leading to Permanent Discontinuation of Study Treatment or Withdrawal from Study by System Organ Class and Preferred Term /by Overall Frequency – Part 2 | IDSL | SAC [1] |
| Laborat | ory: Chemistry | I | | | |

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.17. | Safety | LB17 | Summary of Worst Case Chemistry Results to Potential Clinical Importance (PCI) Criteria Post-Baseline Relative to Baseline – Part 1 | ICH E3 | SAC [1] |
| 3.18. | Safety | LB17 | Summary of Worst Case Chemistry Results to Potential Clinical Importance (PCI) Criteria Post-Baseline Relative to Baseline – Part 2 | ICH E3 | SAC [1] |
| 3.19. | Safety | LB1 | Summary of Chemistry Changes from Baseline – Part 1 | ICH E3 Includes Baseline values | SAC [1] |
| 3.20. | Safety | LB1 | Summary of Chemistry Changes from Baseline – Part 2 | ICH E3<br>Includes Baseline values | SAC [1] |
| Labora | tory: Hematolo | gy | | | |
| 3.21. | Safety | LB17 | Summary of Worst Case Hematology Results to Potential Clinical Importance (PCI) Criteria Post-Baseline Relative to Baseline – Part 1 | ICH E3 | SAC [1] |
| 3.22. | Safety | LB17 | Summary of Worst Case Hematology Results to Potential Clinical Importance (PCI) Criteria Post-Baseline Relative to Baseline – Part 2 | ICH E3 | SAC [1] |
| 3.23. | Safety | LB1 | Summary of Hematology Changes from Baseline – Part 1 | ICH E3 Includes Baseline values. | SAC [1] |
| 3.24. | Safety | LB1 | Summary of Hematology Changes from Baseline – Part 2 | ICH E3<br>Includes Baseline values. | SAC [1] |
| Labora | tory: Urinalysis | 3 | | | |
| 3.25. | Safety | LB15 | Summary of Worst Case Urine Data Results Relative to Normal Range Criteria Post-Baseline Relative to Baseline – Part 1 | ICH E3 | SAC [1] |

| Safety: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.26. | Safety | LB15 | Summary of Worst Case Urine Data Results Relative to Normal Range Criteria Post-Baseline Relative to Baseline – Part 2 | ICH E3 | SAC [1] |
| 3.27. | Safety | LB1 | Summary of Urine Changes from Baseline – Part 1 | ICH E3<br>Includes Baseline values. | SAC [1] |
| 3.28. | Safety | LB1 | Summary of Urine Changes from Baseline– Part 2 | ICH E3<br>Includes Baseline values. | SAC [1] |
| Labora | tory: Abnormal | ities | | | |
| 3.29. | Safety | LB1 | Summary of Grade 1 or Higher Lab Abnormalities– Part 1 | Summary of Treatment Emergent Lab toxicity only. | SAC [1] |
| 3.30. | Safety | LB1 | Summary of Grade 1 or Higher Lab Abnormalities – Part 2 | Summary of Treatment Emergent Lab toxicity only. | SAC [1] |
| Labora | tory: Hepatobil | iary (Liver) | | | |
| 3.31. | Safety | LIVER1 | Summary of Liver Monitoring/Stopping Event Reporting – Part 1 | IDSL | SAC [1] |
| 3.32. | Safety | LIVER1 | Summary of Liver Monitoring/Stopping Event Reporting – Part 1 | IDSL | SAC [1] |
| 3.33. | Safety | LIVER10 | Summary of Subjects Meeting Emergent Hepatobiliary Laboratory Abnormalities Event Reporting – Part 1 | IDSL | SAC [1] |
| 3.34. | Safety | LIVER10 | Summary of Subjects Meeting Emergent Hepatobiliary<br>Laboratory Abnormalities Event Reporting – Part 2 | IDSL | SAC [1] |
| ECG | | | | | |
| 3.35. | Safety | EG1 | Summary of ECG Findings –Part 1 | IDSL Use ECG findings categories (and change from baseline categories, if applicable). | SAC [1] |

| Safety: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.36. | Safety | EG1 | Summary of ECG Findings –Part 2 | IDSL Use ECG findings categories (and change from baseline categories, if applicable). | SAC [1] |
| 3.37. | Safety | EG2 | Summary of Change from Baseline in ECG Values–Part 1 | IDSL<br>Includes Baseline values. | SAC [1] |
| 3.38. | Safety | EG2 | Summary of Change from Baseline in ECG Values–Part 2 | IDSL<br>Includes Baseline values. | SAC [1] |
| 3.39. | Safety | EG1 | Summary of Category of QTc Data–Part 1 | IDSL | SAC [1] |
| 3.40. | Safety | EG1 | Summary of Category of QTc Data-Part 2 | IDSL | SAC [1] |
| 3.41. | Safety | EG1 | Summary of Category of QTc Change from Baseline–Part 1 | IDSL<br>Includes Baseline values. | SAC [1] |
| 3.42. | Safety | EG1 | Summary of Category of QTc Change from Baseline –Part 2 | IDSL<br>Includes Baseline values. | SAC [1] |
| Vital Si | gns | | | | |
| 3.43. | Safety | VS1 | Summary of Vital Signs – Part 1 | ICH E3 | SAC [1] |
| 3.44. | Safety | VS1 | Summary of Vital Signs – Part 2 | ICH E3 | SAC [1] |
| 3.45. | Safety | VS1 | Summary of Change from Baseline in Vital Signs – Part 1 | ICH E3<br>Includes Baseline values. | SAC [1] |
| 3.46. | Safety | VS1 | Summary of Change from Baseline in Vital Signs – Part 2 | ICH E3 Includes Baseline values. | SAC [1] |

### 14.12.8 Safety Figures

| Safety | Safety : Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Labora | tory Values | | | | |
| 3.1. | Safety | As EG9 | Plot of Selected Clinical Lab Tests Mean Change from Baseline by Treatment and Time – Part 1 | Only include scheduled visits and for selected lab test (BNP, Tnp1, ALT, AST, Bili) Plots will be presented with treatment groups overlaid | SAC [1] |
| 3.2. | Safety | As EG9 | Plot of Selected Clinical Lab Tests Mean Change from Baseline by Treatment and Time – Part 2 | Only include scheduled visits and for selected lab test (BNP, Tnp1, ALT, AST, Bili) Plots will be presented with treatment groups overlaid | SAC [1] |
| ECG | | | | · | |
| 3.3. | Safety | EG9 | Plot of Mean Change from Baseline QTcB and QTcF Data by Treatment and Time – Part 1 | Plots will be presented with treatment groups overlaid | SAC [1] |
| 3.4. | Safety | EG9 | Plot of Mean Change from Baseline QTcB and QTcF Data by Treatment and Time – Part 2 | Plots will be presented with treatment groups overlaid | SAC [1] |
| Vital Si | gns | | | | |
| 3.5. | Safety | As EG8 | Box Plot of Change from Baseline for Vital Signs by Treatment and Time – Part 1 | Plots will be presented with treatment groups overlaid | SAC [1] |
| 3.6. | Safety | As EG8 | Box Plot of Change from Baseline for Vital Signs by Treatment and Time – Part 2 | Plots will be presented with treatment groups overlaid | SAC [1] |

### 14.12.9 Pharmacokinetic Tables

| Pharma | Pharmacokinetic: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Pharma | acokinetic | | | | |
| 5.1. | PK | PK14 | Listing of Derived Plasma GSK2838232 PK Parameters – Part 1A | Sort by participant and treatment | SAC [1] |
| 5.2. | PK | PK14 | Listing of Derived Plasma GSK2838232 PK Parameters – Part 1B | Sort by participant and treatment | SAC [1] |
| 5.3. | PK | PK13 | Listing of Derived Plasma GSK2838232 PK Parameters – Part 2 | Sort by participant and treatment | SAC [1] |
| Bioava | ilability | | | | |
| 5.4. | PK | PK01 | Summary Statistics of Plasma GSK2838232 PK Concentration-<br>Time Data, Bioavailability | | SAC [1] |
| 5.5. | PK | PK04 | Summary Statistics of Derived Plasma GSK2838232 PK Parameters by Treatment, Bioavailability | | SAC [1] |
| 5.6. | PK | PK05 | Summary Statistics of Log <sub>e</sub> -transformed Derived Plasma GSK2838232 PK Parameters, Bioavailability | | SAC [1] |
| 5.7. | PK | Non-Standard1 | Summary of Result of Plasma GSK2838232 PK Parameter<br>Treatment Comparisons for Relative Bioavailability | | SAC [1] |
| 5.8. | PK | PK15 | Listing of Individual Derived Plasma GSK2838232 PK Parameters Treatment Ratios | PK Parameter: AUC(0-inf), and Cmax<br>Ratio: Tablet/Capsule | SAC [1] |
| Food E | ffect | | | , | |
| 5.9. | PK | PK01 | Summary Statistics of Plasma GSK2838232 PK Concentration-<br>Time Data, Food Effect | | SAC [1] |
| 5.10. | PK | PK04 | Summary Statistics of Derived Plasma GSK2838232 PK Parameters by Treatment, Food Effect | | SAC [1] |

| Pharma | Pharmacokinetic: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 5.11. | PK | PK05 | Summary Statistics of Log <sub>e</sub> -transformed Derived Plasma GSK2838232 PK Parameters, Food Effect | | SAC [1] |
| 5.12. | PK | Non-Standard2 | Summary of Result of Plasma GSK2838232 PK Parameter Treatment Comparisons for Food Effect | | SAC [1] |
| 5.13. | PK | PK15 | Listing of Individual Derived Plasma GSK2838232 PK<br>Parameters Treatment Ratios | PK Parameter: AUC(0-inf), Cmax, and tmax Ratio: Fed/Fasted | SAC [1] |
| Steady | State Assessm | nents and Accumu | ılation | | |
| 5.14. | PK | PK04 | Summary Statistics of Plasma GSK2838232 PK Parameters by Treatment and by Day – Part 2 | Day 1 & Day 11 | SAC [1] |
| 5.15. | PK | PK04 | Summary Statistics of Derived Plasma GSK2838232 PK Parameters by Treatment and by Day – Part 2 | Day 1 & Day 11 | SAC [1] |
| 5.16. | PK | PK05 | Summary of Log <sub>e</sub> -transformed Derived Plasma GSK2838232 PK Parameters by Treatment and by Day – Part 2 | Day 1 & Day 11 | SAC [1] |
| 5.17. | PK | Non-Standard3 | Summary of Results of GSK2838232 PK Parameter Treatment Comparisons -Accumulation Assessments- Part 2 | One for each treatment | SAC [1] |
| 5.18. | PK | Non-Standard4 | Summary Results of Steady State GSK2838232 Concentrations<br>Assessments- Part 2 | One for each treatment | SAC [1] |

### 14.12.10 Pharmacokinetic Figures

| Pharmacokinetic : Figures | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Biovail | ability | | | | |
| 5.1. | PK | PK16B | Individual Plasma GSK2838232 PK Concentration-Time Plots for Relative Bioavailability | Linear and Semi-Log Scale By participant, overlay all treatments for each participant | SAC [1] |
| 5.2. | PK | PK17 | Mean Plasma GSK2838232 PK Concentration for Relative Bioavailability | Linear and Semi-Log Scale Overlay all treatments | SAC [1] |
| 5.3. | PK | PK18 | Median Plasma GSK2838232 PK Concentration for Relative Bioavailability | Linear and Semi-Log Scale<br>Overlay all treatments | SAC [1] |
| 5.4. | PK | PK28 | Geometric Mean Treatment Ratio and 90% Confidence Interval of GSK2838232 PK Parameter for the Relative Bioavailability | | SAC [1] |
| 5.5. | PK | PK25 | Comparative Plot of Individual Plasma GSK2838232 PK Parameters for Relative Bioavailability by treatment | | SAC [1] |
| Food E | ffect | | | | |
| 5.6. | PK | PK16A | Individual Plasma GSK2838232 PK Concentration-Time Plots for Food Effect | Linear and Semi-Log Scale By participant, overlay all treatments for each participant | SAC [1] |
| 5.7. | PK | PK17 | Mean Plasma GSK2838232 PK Concentration for Food Effect | Linear and Semi-Log Scale Overlay all treatments | SAC [1] |
| 5.8. | PK | PK18 | Median Plasma GSK2838232 PK Concentration for Food Effect | Linear and Semi-Log Scale Overlay all treatments | SAC [1] |
| 5.9. | PK | PK28 | Geometric Mean Treatment Ratio and 90% Confidence Interval of GSK2838232 PK Parameter for Food Effect | | SAC [1] |

| Pharma | cokinetic : Fig | ures | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 5.10. | PK | PK25 | Comparative Plot of Individual Plasma GSK2838232 PK Parameters for Food Effect by treatment | | SAC [1] |
| Steady | State Assessm | nents and Accum | ulation | | |
| 5.11. | PK | PK16a | Individual Plasma GSK2838232 PK Concentration-Time Plots by Day – Part 2 | Linear and Semi-Log Scale By participant, overlay days for each participant | SAC [1] |
| 5.12. | PK | PK17 | Mean Plasma GSK2838232 PK Concentration by Day – Part 2 | Linear and Semi-Log Scale | SAC [1] |
| 5.13. | PK | PK18 | Median Plasma GSK2838232 PK Concentration by Day – Part 2 | Linear and Semi-Log Scale | SAC [1] |
| 5.19. | PK | PK16a | Individual Plasma GSK2838232 Predose Concentration-Time Plots for Steady State Assessment – Part 2 | Linear and Semi-Log Scale Overlay all individual profile with all days profiles | SAC [1] |
| 5.20. | PK | PK17 | Mean Plasma GSK2838232 Concentration-Time Plots for Steady State Assessment – Part 2 | Linear and Semi-Log Scale | SAC [1] |
| 5.21. | PK | PK18 | Median Plasma GSK2838232 Concentration-Time Plots for Steady State Assessment – Part 2 | Linear and Semi-Log Scale | SAC [1] |
| 5.22. | PK | PK16a | Individual and Box Plot of Plasma GSK2838232 PK Parameters by Day – Part 2 | Include all the PK parameters. | SAC [1] |
| 5.23. | PK | PK25 | Comparative Plot of Plasma GSK2838232 PK Parameters for Accumulation | Linear and Log Scale | SAC [1] |

### 14.12.11 Pharmacokinetic Population (PopPK) Tables

Not applicable.

### 14.12.12 Pharmacokinetic Population (PopPK) Figures

Not applicable.

### 14.12.13 Pharmacodynamic Tables

Not applicable.

### 14.12.14 Pharmacodynamic Figures

Not applicable.

### 14.12.15 Pharmacokinetic / Pharmacodynamic Tables

Not applicable.

### 14.12.16 Pharmacokinetic / Pharmacodynamic figures

Not applicable.

### **14.12.17 ICH Listings**

| ICH: Lis | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Particip | oant Dispositio | n | | | |
| 1. | Screened | ES7 | Listing of Reasons for Screen Failure – Part 1 | Journal Guidelines | SAC [1] |
| 2. | Screened | ES7 | Listing of Reasons for Screen Failure – Part 2 | Journal Guidelines | SAC [1] |
| 3. | Safety | ES3 | Listing of Reasons for Study Withdrawal – Part 1 | ICH E3 | SAC [1] |
| 4. | Safety | ES2 | Listing of Reasons for Study Withdrawal – Part 2 | ICH E3 | SAC [1] |
| 5. | Safety | SD3 | Listing of Reasons for Study Treatment Discontinuation – Part 1 | ICH E3 | SAC [1] |
| 6. | Safety | SD2 | Listing of Reasons for Study Treatment Discontinuation – Part 2 | ICH E3 | SAC [1] |
| 7. | Safety | BL1 | Listing of Participants for Whom the Treatment Blind was Broken – Part 2 | ICH E3 | SAC [1] |
| 8. | Safety | CP_RA1x | Listing of Planned and Actual Treatments – Part 1 | IDSL | SAC [1] |
| 9. | Safety | CP_RA1p | Listing of Planned and Actual Treatments – Part 2 | IDSL | SAC [1] |
| Protoco | ol Deviations | | | | • |
| 10. | Safety | DV2A | Listing of Important Protocol Deviations – Part 1 | ICH E3 Listing also includes analysis population exclusions. | SAC [1] |
| 11. | Safety | DV2 | Listing of Important Protocol Deviations – Part 2 | ICH E3 Listing also includes analysis population exclusions. | SAC [1] |
| 12. | Safety | IE4 | Listing of Participants with Inclusion/Exclusion Criteria Deviations – Part 1 | ICH E3 | SAC [1] |
| 13. | Safety | IE3 | Listing of Participants with Inclusion/Exclusion Criteria Deviations – Part 2 | ICH E3 | SAC [1] |

| ICH: Li | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Popula | tions Analysed | | | | |
| 14. | Safety | SP3A | Listing of Participants Excluded from Any Population – Part 1 | ICH E3 | SAC [1] |
| 15. | Safety | SP3 | Listing of Participants Excluded from Any Population – Part 2 | ICH E3 | SAC [1] |
| Demog | raphic and Bas | eline Characteris | tics | | |
| 16. | Safety | DM4 | Listing of Demographic Characteristics – Part 1 | ICH E3 | SAC [1] |
| 17. | Safety | DM2 | Listing of Demographic Characteristics – Part 2 | ICH E3 | SAC [1] |
| 18. | Safety | DM10 | Listing of Race – Part 1 | ICH E3 | SAC [1] |
| 19. | Safety | DM9 | Listing of Race – Part 2 | ICH E3 | SAC [1] |
| Prior a | nd Concomitan | t Medications | | | |
| 20. | Safety | CP_CM4 | Listing of Concomitant Medications – Part 1 | IDSL | SAC [1] |
| 21. | Safety | CP_CM3 | Listing of Concomitant Medications – Part 2 | IDSL | SAC [1] |
| Exposi | ure and Treatme | ent Compliance | | | |
| 22. | Safety | EX4 | Listing of Exposure Data – Part 1 | ICH E3 | SAC [1] |
| 23. | Safety | EX3 | Listing of Exposure Data – Part 2 | ICH E3 | SAC [1] |
| Advers | e Events | | | | |
| 24. | Safety | CP_AE9 | Listing of All Adverse Events – Part 1 | ICH E3 | SAC [1] |
| 25. | Safety | CP_AE8 | Listing of All Adverse Events – Part 2 | ICH E3 | SAC [1] |
| 26. | Safety | AE7 | Listing of Participant Numbers for Individual Adverse Events – Part 1 | ICH E3 | SAC [1] |
| 27. | Safety | AE7 | Listing of Participant Numbers for Individual Adverse Events – Part 2 | ICH E3 | SAC [1] |
| 28. | Safety | AE2 | Listing of Relationship Between Adverse Event System Organ Classes, Preferred Terms, and Verbatim Text – Part 1 | IDSL | SAC [1] |

| ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 29. | Safety | AE2 | Listing of Relationship Between Adverse Event System Organ Classes, Preferred Terms, and Verbatim Text – Part 2 | IDSL | SAC [1] |
| Serious | and Other Sig | nificant Adverse l | Events | | • |
| 30. | Safety | CP_AE9a | Listing of Fatal Serious Adverse Events – Part 1 | ICH E3 | SAC [1] |
| 31. | Safety | CP_AE8a | Listing of Fatal Serious Adverse Events – Part 2 | ICH E3 | SAC [1] |
| 32. | Safety | CP_AE9a | Listing of Non-Fatal Serious Adverse Events – Part 1 | ICH E3 | SAC [1] |
| 33. | Safety | CP_AE8a | Listing of Non-Fatal Serious Adverse Events – Part 2 | ICH E3 | SAC [1] |
| 34. | Safety | AE14 | Listing of Reasons for Considering as a Serious Adverse Event | ICH E3 | SAC [1] |
| 35. | Safety | CP_AE9a | Listing of Adverse Events Leading to Withdrawal from Study / Permanent Discontinuation of Study Treatment – Part 1 | ICH E3 | SAC [1] |
| 36. | Safety | CP_AE8a | Listing of Adverse Events Leading to Withdrawal from Study / Permanent Discontinuation of Study Treatment – Part 2 | ICH E3 | SAC [1] |
| 37. | Safety | CP_AE9a | Listing of Grade 3 or 4 Adverse Events – Part 1 | Division of AIDS Table For Grading | SAC [1] |
| 38. | Safety | CP_AE8a | Listing of Grade 3 or 4 Adverse Events – Part 2 | Division of AIDS Table For Grading | SAC [1] |
| Hepato | biliary (Liver) | | | | |
| 39. | Safety | MH2 | Listing of Medical Conditions for Participants with Liver Stopping<br>Events – Part 1 | IDSL | SAC [1] |
| 40. | Safety | MH2 | Listing of Medical Conditions for Participants with Liver Stopping Events – Part 2 | IDSL | SAC [1] |
| 41. | Safety | SU2 | Listing of Substance Use for Participants with Liver Stopping Events – Part 1 | IDSL | SAC [1] |
| 42. | Safety | SU2 | Listing of Substance Use for Participants with Liver Stopping Events – Part 2 | IDSL | SAC [1] |
| All Lab | oratory | | | · | |

| ICH: Lis | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 43. | Safety | LB13 | Listing of Reference Ranges for Clinical Laboratory Tests | | SAC [1] |
| 44. | Safety | LB6 | Listing of Hematology Data– Part 1 | If any laboratory test results are outside of the reference range, they will be flagged with high/low and/or toxicity grade in the listing | SAC [1] |
| 45. | Safety | LB5 | Listing of Hematology Data– Part 2 | If any laboratory test results are outside of the reference range, they will be flagged with high/low and/or toxicity grade in the listing | SAC [1] |
| 46. | Safety | LB6 | Listing of Clinical Chemistry Data- Part 1 | If any laboratory test results are outside of the reference range, they will be flagged with high/low and/or toxicity grade in the listing | SAC [1] |
| 47. | Safety | LB5 | Listing of Clinical Chemistry Data- Part 2 | If any laboratory test results are outside of the reference range, they will be flagged with high/low and/or toxicity grade in the listing | SAC [1] |
| 48. | Safety | LB6 | Listing of Urinalysis Data– Part 1 | If any laboratory test results are outside of the reference range, they will be flagged with high/low and/or toxicity grade in the listing | SAC [1] |
| 49. | Safety | LB5 | Listing of Urinalysis Data– Part 2 | If any laboratory test results are outside of the reference range, they will be flagged with high/low and/or toxicity grade in the listing | SAC [1] |

| ICH: Listings | | | | | | |
|---|---|---|---|---|---|--|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] | |
| 50. | Safety | LB6 | Listing of All Laboratory Data for Participants with Any Value of Potential Clinical Importance– Part 1 | ICH E3 May be split into separate listings by chemistry, hematology, etc. Display ALL labs for a participant who experienced a value of potential clinical importance. | SAC [1] | |
| 51. | Safety | LB5 | Listing of All Laboratory Data for Participants with Any Value of Potential Clinical Importance– Part 2 | ICH E3 May be split into separate listings by chemistry, hematology, etc. Display ALL labs for a participant who experienced a value of potential clinical importance. | SAC [1] | |
| 52. | Safety | LB6 | Listing of Lab Results Identified as Adverse Events– Part 1 | Lab results identified as AEs. Only needed if there are a sufficient number of labs identified as AEs. | SAC [1] | |
| 53. | Safety | LB5 | Listing of Lab Results Identified as Adverse Events – Part 2 | Lab results identified as AEs. Only needed if there are a sufficient number of labs identified as AEs. | SAC [1] | |
| 54. | Safety | LB6 | Listing of Grade 2 or Higher Lab Abnormalities – Part 1 | | SAC [1] | |
| 55. | Safety | LB5 | Listing of Grade 2 or Higher Lab Abnormalities – Part 2 | | SAC [1] | |
| 56. | Safety | LB14 | Listing of Laboratory Data with Character Results – Part 1 | ICH E3 | SAC [1] | |
| 57. | Safety | LB14 | Listing of Laboratory Data with Character Results – Part 2 | ICH E3 | SAC [1] | |
| 58. | Safety | UR2B | Listing of Urinalysis Data for Participants with Any Value of Potential Clinical Importance – Part 1 | ICH E3 Display ALL data for a participant who experienced a value of potential clinical importance. | SAC [1] | |
| ICH: Lis | ICH: Listings | | | | | | |
|---|---|---|---|---|---|--|--|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] | | |
| 59. | Safety | UR2A | Listing of Urinalysis Data for Participants with Any Value of Potential Clinical Importance – Part 2 | ICH E3 Display ALL data for a participant who experienced a value of potential clinical importance. | SAC [1] | | |
| ECG and | d Holter | | | | | | |
| 60. | Safety | EG4 | Listing of All ECG Values for Participants with Any Value of Potential Clinical Importance – Part 1 | IDSL | SAC [1] | | |
| 61. | Safety | EG3 | Listing of All ECG Values for Participants with Any Value of Potential Clinical Importance – Part 2 | IDSL | SAC [1] | | |
| 62. | Safety | EG6 | Listing of All ECG Findings for Participants with an Abnormal ECG Finding – Part 1 | IDSL | SAC [1] | | |
| 63. | Safety | EG5 | Listing of All ECG Findings for Participants with an Abnormal ECG Finding – Part 2 | IDSL | SAC [1] | | |
| 64. | Safety | HM8 | Listing of Holter Monitoring – Part 1 | IDSL | SAC [1] | | |
| 65. | Safety | HM8 | Listing of Holter Monitoring – Part 2 | IDSL | SAC [1] | | |
| Vital Sig | ns | | | | | | |
| 66. | Safety | VS5 | Listing of All Vital Signs Data for Participants with Any Value of Potential Clinical Importance – Part 1 | IDSL | SAC [1] | | |
| 67. | Safety | VS4 | Listing of All Vital Signs Data for Participants with Any Value of Potential Clinical Importance – Part 2 | IDSL | SAC [1] | | |

# 14.12.18 Non-ICH Listings

| Non-IC | H: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Pharma | cokinetic | | | | |
| 68. | PK | PK08 | Listing of Plasma GSK2838232 PK Concentration-Time Data – Part 1A | Sort by participant, treatment, day, and time | SAC [1] |
| 69. | PK | PK08 | Listing of Plasma GSK2838232 PK Concentration-Time Data – Part 1B | Sort by participant, treatment, day, and time | SAC [1] |
| 70. | PK | PK07 | Listing of Plasma GSK2838232 PK Concentration-Time Data – Part 2 | Sort by participant, treatment, day, and time | SAC [1] |
| PK Stat | PK Statistical Analysis | | | | |
| 71. | PK | SAS output of<br>Table5.6 | SAS Output of Summary Results of GSK2838232 PK Parameter Treatment Comparisons for the Relative Bioavailability – Part 1A | | SAC [1] |
| 72. | PK | SAS output of<br>Table 5.10 | SAS Output of Summary Results of GSK2838232 PK Parameter Treatment Comparisons for the Food Effect – Part 1B | | SAC [1] |
| 73. | PK | SAS output of<br>Table 5.16 | SAS Output of Summary Results of Steady-State GSK2838232<br>Concentrations Assessment – Part 2 | | SAC [1] |
| 74. | PK | SAS output of Table 5.17 | SAS Output of Summary Results of GSK2838232 PK Parameter Treatment Comparisons – Accumulation Ratio – Part 2 | | SAC [1] |

# 14.13 Appendix 13: Example Mock Shells for Data Displays


Protocol: XXXXXX 

Population: PK Parameter

#### Geometric LSMean 90% Confidence Interval Comparison PK Parameter Test/Ref. (N=12)(N=12)Ratio CVw (%) AUC (0-inf) (h\*ng/mL) G vs A 1029.925 1469.603 1.4269 (1.1962,1.7021) 24.18 AUC (0-t) (h\*ng/mL)989.181 1443.028 1.4588 (1.2320,1.7274) 23.14 G vs A AUC (0-24) (h\*ng/mL)G vs A 460.663 681.540 1.4795 (1.2479,1.7541) 23.32 Cmax (ng/mL) G vs A 30.126 47.561 1.5787 (1.3118,1.9000) 25.43 21.782 1.4161 (1.2044,1.6649) 22.14 C24 (ng/mL) G vs A 15.382 t1/2 (h) G vs A 19.770 18.779 0.9499 (0.8578,1.0519) 13.85

A: Treatment description G:Treatment description


205820


> Protocol: XXXXXX Population: PK Parameter 

Table X.XX
Summary Results of Treatment Comparisons for the Food Effect - Part 1B

#### Geometric LSMean

| PK Parameter | Comparison<br>Test/Ref. | G<br>(N=12) | F<br>(N=11) | Ratio | 90% Confidence<br>Interval | CVw (%) |
|---|---|---|---|---|---|---|
| AUC (0-inf) (h*ng/mL) | F (Fed) Vs G (Fasted | 1) 1469.603 | 2327.794 | | (1.4120,1.7768) | |
| AUC $(0-t)$ $(h*ng/mL)$ | F (Fed) Vs G (Fasted | 1) 1443.028 | 2299.310 | 1.5934 | (1.4185,1.7899) | 15.13 |
| AUC $(0-24)$ $(h*ng/mL)$ | F (Fed) Vs G (Fasted | 681.540 | 1048.089 | 1.5378 | (1.3761,1.7185) | 14.50 |
| Cmax (ng/mL) | F (Fed) Vs G (Fasted | 47.561 | 77.132 | 1.6217 | (1.3762,1.9111) | 21.81 |
| C24 (ng/mL) | F (Fed) Vs G (Fasted | 1) 21.782 | 35.718 | 1.6398 | (1.4417,1.8653) | 16.80 |
| t1/2 (h) | F (Fed) Vs G (Faster | 18 779 | 18 582 | 0 9895 | (0.9155-1.0695) | 10 14 |

G: GSKXXXXXX Capsule 100mg + XXX F: GSKXXXXXX Capsule 100mg + Food + XXX


205820

Page 1 of n Example: Non-Standard3

> Protocol: XXXXXX Population: PK Parameter 

Table X.XX
Summary Results of GSK XXXXXXX PK Parameter Treatment Comparisons - Accumulation Ratio - Part 2

| | | Treatment | Comp<br>Tes | | | | | _Geometri<br>Ref. | c LSmean_<br>Test. | Ratio | 90% Confidence<br>Interval | CVb(%) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Accumulation<br>AUC(0-tau) | Ratio | RD20mg+RTV | Day | 11 | vs | Day | 1 | 175.060 | 449.021 | 2.5650 | (1.9931,3.3008) | 21.94 |
| | | RD50mg+RTV | Day | 11 | VS | Day | 1 | 265.413 | 1087.465 | 4.0973 | (2.7102, 6.1943) | 36.68 |
| | | CapRD100mg+RTV | | | | Day | | 635.446 | 2411.467 | 3.7949 | (2.8185, 5.1096) | 25.99 |
| | | CapRD200mg+RTV | | | | Day | | 1056.386 | 4014.085 | 3.7998 | (3.1234, 4.6227) | 16.97 |
| | | CapRDQ12H200mg | | | | Day | | 267.134 | 742.180 | 2.7783 | (2.3991, 3.2175) | 12.67 |
| Accumulation<br>Cmax | Ratio | RD20mg+RTV | Day | 11 | VS | Day | 1 | 11.109 | 25.335 | 2.2807 | (1.6717,3.1114) | 27.18 |
| | | RD50mg+RTV | Day | 11 | VS | Day | 1 | 17.098 | 56.614 | 3.3111 | (2.2479.4.8771) | 34.23 |
| | | CapRD100mg+RTV | | | | Day | | 46.172 | 129.785 | 2.8109 | (2.0427, 3.8681) | 27.97 |
| | | CapRD200mg+RTV | | | | Day | | 75.033 | 224.886 | 2.9972 | (2.4531, 3.6619) | 17.35 |
| | | CapRDQ12H200mg | | | | Day | | 51.237 | 96.085 | 1.8753 | (1.6520,2.1288) | 10.93 |
| Accumulation<br>Ctau | Ratio | RD20mg+RTV | Day | 11 | VS | Day | 1 | 5.673 | 14.525 | 2.5604 | (2.0159, 3.2521) | 20.77 |
| CLau | | RD50mg+RTV | Day | 11 | VS | Dav | 1 | 8.919 | 37.403 | 4.1939 | (2.8754, 6.1169) | 33.31 |
| | | CapRD100mg+RTV | | | | Day | | 20.560 | 78.196 | 3.8033 | (2.6625, 5.4329) | 31.39 |
| | | CapRD200mg+RTV | | | | Day | | 36.696 | 136.681 | 3.7247 | (2.9585, 4.6892) | 19.99 |
| | | CapRD012H200mg | | | | Day | | 18.364 | 39.144 | 2.1315 | (1.7403, 2.6107) | 17.56 |
| | | caphogizhzoulig | Day | 11 | 42 | Day | 1 | TO. 204 | 22.144 | 2.1313 | (1.1400,2.0101) | 11.00 |


205820


Protocol: XXXXXX Page 1 of 2 Population: PK Parameter

Table X.XX

Summary Results of Steady-State GSKXXXXXXX Concentrations Assessment - Part 2

| Included<br>Days | Treatment | Slope | 90% Confidence<br>Interval |
|---|---|---|---|
| Days 3-11 | RD20mg+RTV | 0.023 | (0.009,0.037) |
| | RD50mg+RTV | 0.082 | (0.065,0.100) |
| | CapRD100mg+RTV | 0.058 | (0.044,0.072) |
| | CapRD200mg+RTV | 0.033 | (0.018,0.047) |
| | CapRD212H200mg | 0.007 | (-0.005,0.019) |
| Days 4-11 | RD20mg+RTV | 0.006 | (-0.009,0.020) |
| | RD50mg+RTV | 0.063 | (0.046,0.081) |
| | CapRD100mg+RTV | 0.037 | (0.022,0.051) |
| | CapRD200mg+RTV | 0.003 | (-0.008,0.015) |
| | CapRDQ12H200mg | 0.004 | (-0.010,0.018) |
| Days 5-11 | RD20mg+RTV | -0.012 | (-0.029,0.005) |
| | RD50mg+RTV | 0.038 | (0.022,0.053) |
| | CapRD100mg+RTV | 0.013 | (-0.001,0.027) |
| | CapRD200mg+RTV | -0.004 | (-0.018,0.010) |
| | CapRDQ12H200mg | 0.001 | (-0.019,0.020) |
| Days 6-11 | RD20mg+RTV<br>RD50mg+RTV<br>CapRD100mg+RTV<br>CapRD200mg+RTV | -0.021<br>0.029<br>0.008<br>-0.009 | (-0.041,-0.001)<br>(0.010,0.048)<br>(-0.011,0.028)<br>(-0.027,0.009)<br>(-0.022,0.025) |

# PAREXEL International Statistical Analysis Plan Addendum

## STATISTICAL ANALYSIS PLAN ADDENDUM

#### 205820

Reporting and Analysis Plan for: A Two Part Study to Assess i) the Relative Bioavailability and Food Effect of a Novel Tablet Formulation of Boosted-GSK2838232 Compared to Capsule and ii) the Safety and Pharmacokinetics of Repeated Once-Daily Doses of Non boosted GSK2838232

Version: Final 1.0

Date: 16/Apr/2018

GlaxoSmithKline Research & Development Limited 205820

Final 1.0

16/Apr/2018

# Statistical Analysis Plan Addendum

### **REVISION HISTORY**

| Version | Version Date | Author | <b>Summary of Changes Made</b> |
|-----------|--------------|--------|--------------------------------|
| Final 1.0 | See Footer | PPD | New Document |

GlaxoSmithKline Research & Development Limited 205820

Final 1.0

16/Apr/2018

# Statistical Analysis Plan Addendum

# SIGNATURE PAGE - GLAXOSMITHKLINE RESEARCH & DEVELOPMENT LIMITED

#### **Declaration**

The undersigned has/have reviewed and agree to the statistical analyses and procedures of this clinical study as presented in this document.

| Principal Biostatistician (PCPS, GSK) | Date (DD Mmm YY) |
|----------------------------------------------------|------------------|
| PPD Director, Clinical Pharmacology (CPMS, GSK) | Date (DD Mmm YY) |
| PPD | Date (DD Mmm YY) |
| Principal Clinical Research Scientist (CPSSO, GSK) | |
| PPD (CRAN) | Date (DD Mmm YY) |
| Sm Executive Medical Director (GSK) | |

GlaxoSmithKline Research & Development Limited 205820

Final 1.0

16/Apr/2018

TP-EP.BS-WW-008-04 Effective date: 29 Jul 15

Related to: SOP-EP.BS-WW-002 Page 3 of 47

# PAREXEL International Statistical Analysis Plan Addendum

| PPD | Date (DD Mmm YY) |
|--------------------------------------------|------------------|
| Principal Programmer (PCPS, GSK) | |
| PPD | Date (DD Mmm YY) |
| Principal Data Manager (CPSSO, GSK) | |
| PPD | Date (DD Mmm YY) |
| Senior Director, Biostatistics (PCPS, GSK) | |
| PPD | Date (DD Mmm YY) |
| Manager, Programming (PCPS, GSK) | |

GlaxoSmithKline Research & Development Limited 205820

Final 1.0

16/Apr/2018

# Statistical Analysis Plan Addendum

## **SIGNATURE PAGE - PAREXEL**

### **Declaration**

| The undersigned agree to the statistical analyses and procedures of this clinical study. | |
|---|---|
| If this document has been signed electronically, signature(s) and date(s) are present at the end of the document: | |
| Document prepared and approved by: | |
| PPD | Date (DD Mmm YY) |
| Sr. Biostatistician | |
| Document prepared and approved by: | |
| PPD | Date (DD Mmm YY) |
| QCD Senior Scientific | |

GlaxoSmithKline Research & Development Limited 205820

Final 1.0

16/Apr/2018

# Statistical Analysis Plan Addendum

### **TABLE OF CONTENTS**

| REVI | SION H | IISTORY | 2 |
|---|---|---|---|
| SIGN | ATURE | E PAGE - GLAXOSMITHKLINE RESEARCH & DEVELOPMENT LIMITED. | 3 |
| SIGN | ATURE | E PAGE - PAREXEL | 5 |
| TABI | LE OF C | CONTENTS | 6 |
| LIST | OF TAI | BLES | 7 |
| ABBI | REVIAT | TION AND ACRONYM LIST | 8 |
| 1. | STA | ΓISTICAL ANALYSIS PLAN ADDENDUM | 9 |
| 2. | OVE | RVIEW OF CHANGES REQUIRED | . 10 |
| | 2.1 | Summary of Changes | . 10 |
| | 2.2 | Study objective and secondary end point | . 11 |
| | 2.3 | Study Design | . 11 |
| | 2.4 | Statistical Hypothesis/Statistical Analysis | . 11 |
| | 2.5 | Study Treatment and Sub-group Display Descriptors | . 11 |
| | 2.6 | Concomitant Medications | . 13 |
| | 2.7 | Treatment Compliance and Protocol Deviations | . 13 |
| | 2.8 | Derived Pharmacokinetic Parameters | . 13 |
| | 2.9 | Statistical Analysis/Method | . 15 |
| 3. | TAB | LES/LISTINGS/FIGURES | . 16 |
| | 3.1 | Final Tables, Listings and Figures | . 16 |
| 4. | SHEI | LLS | . 45 |
| 5. | REFI | ERENCES | . 47 |

GlaxoSmithKline Research & Development Limited 205820

Final 1.0

16/Apr/2018

# Statistical Analysis Plan Addendum

### LIST OF TABLES

| Table 1 | Study Population Tables | 17 |
|----------|--------------------------------------------|----|
| Table 2 | Safety Tables | 19 |
| Table 3 | Safety Figures | 24 |
| Table 4 | Pharmacokinetic Tables | 25 |
| Table 5 | Pharmacokinetic Figures | 27 |
| Table 6 | ICH Listings | 30 |
| Table 7 | Non-ICH Lisitngs | 36 |
| Table 8 | Study Population Tables (Changes from RAP) | 37 |
| Table 9 | Safety Figures (Changes from RAP) | 38 |
| Table 10 | Pharmacokinetic Tables (Changes from RAP) | 39 |
| Table 11 | Pharmacokinetic Figures (Changes from RAP) | 40 |
| Table 12 | ICH Listing (Changes from RAP) | 43 |
| Table 13 | Non-ICH Listings (Change from RAP) | 44 |

GlaxoSmithKline Research & Development Limited 205820

Final 1.0

16/Apr/2018

# Statistical Analysis Plan Addendum

### ABBREVIATION AND ACRONYM LIST

| Abbreviation / Acronym | Definition / Expansion |
|---|---|
| AUC | Area under the concentration-time curve |
| AUC <sub>(0-inf)</sub> | AUC from time zero extrapolated to infinity |
| $\mathrm{AUC}_{(0\text{-t})}$ | AUC from time zero to the last quantifiable concentration |
| $\mathrm{AUC}_{(0\text{-}	au),\mathrm{ss}}$ | AUC over the dosing interval at steady state |
| BLQ | Below the lower limit of quantification |
| CI | Confidence interval |
| $C_{last}$ | Last quantifiable concentration at t <sub>last</sub> |
| $CL_R$ | Renal clearance |
| CL/F | Apparent clearance following oral administration |
| CL/F,ss | Apparent clearance following oral administration at steady state |
| CSP | Clinical Study Protocol |
| $C_{\text{max}}$ | Maximum observed concentration |
| $C_{\text{min}}$ | Minimum observed concentration in the dosing interval |
| $C_{trough}$ | Concentration immediately prior to dosing |
| CV | Coefficient of variation |
| PK | Pharmacokinetic |
| $R_{ac}$ | Accumulation ratio |
| RAP | Report And Analysis Plan |
| SAP | Statistical Analysis Plan |
| SD | Standard deviation |
| SE | Standard error of the mean |
| $t_{\frac{1}{2}}$ | Apparent terminal elimination half-life |
| $t_{1/2,SS}$ | Apparent terminal elimination half-life at steady state |
| $t_{last}$ | Time of last quantifiable concentration |
| $t_{max}$ | Time corresponding to occurrence of $C_{max}$ |
| $\lambda_{\mathrm{z}}$ | Terminal elimination rate constant |
| $\lambda_{z,ss}$ | Terminal elimination rate constant at steady state |
| %AUC <sub>ex</sub> | Percentage of $AUC_{(0-inf)}$ obtained by extrapolation |
| GlaxoSmithKline Research & | Final 1.0 |
| Development Limited<br>205820 | 16/Apr/2018 |

TP-EP.BS-WW-008-04 Effective date: 29 Jul 15

Related to: SOP-EP.BS-WW-002 Page 8 of 47

### Statistical Analysis Plan Addendum

### 1. STATISTICAL ANALYSIS PLAN ADDENDUM

The Statistical Analysis Plan (SAP) Addendum details the changes and/or additional analyses required that are not currently described in the final RAP Version **1.0** dated 07/Dec/2017. The SAP Addendum describes any deviations from the planned analyses, additional analyses and if applicable, new Tables, Listings and Figures (TLFs) that are to be produced.

As Sponsor (GlaxoSmithKline Research & Development Limited) does not have any template available for RAP Addendum, PAREXEL Template of SAP Addendum is used to document the changes after database lock and finalization of the RAP.

GlaxoSmithKline Research & Development Limited 205820

Final 1.0

16/Apr/2018

### Statistical Analysis Plan Addendum

### 2. OVERVIEW OF CHANGES REQUIRED

#### 2.1 Summary of Changes

- Secondary end point is considered as pre-dose concentration on days 3 to 11 rather than pre-dose concentration on day 2 to 11. This is applicable to final RAP Sections 2.2, 2.4 and 9.2.5
- PK parameter Ctrough is calculated for days 3 to 11 rather than for days 2 to 11. This is applicable to final RAP Sections 9.1.1.2, and 9.2.1.2
  - However Ctrough should not be considered as PK Parameter of the study and this should not be included in ADPP dataset and those values can only be used from ADPC dataset directly and use for Steady State Assessment only. No summary statistics will be provided for this PK parameter.
- Part 2 treatments is changed as Treatment R = GSK2838232 500 mg tablet fed rather than D=GSK2838232 500 mg/r tablet fed and Treatment P=Placebo than Treatment E=Placebo. This is applicable to final RAP Section 2.3
- Listing and summary of the protocol deviation should be presented for all Important Protocol Deviation rather than all Protocol Deviation. This is applicable to final RAP section 6.5.
- For each of the PK parameters given in section of RAP, for the summary statistics calculation, geometric mean associated with 95% CI should be calculated for each treatment group; however in RAP geometric mean associated with 90% CI should be calculated for each treatment group for the summary statistics. This is applicable to RAP sections 9.1.1.2 and 9.2.1.2
- In the statistical methodology, analysis for the steady state assessment should only be mentioned as predose concentrations from days 3 to 11, and no Ctrough or Ctau terminology will be considered for this analysis.

There will be no changes to the structure/format of the tables, figures and listings based on this change. The details of these changes are provided from sections 2.2 to 2.9 below. Details of the changes in the Tables, Listings and Figures are mainly due to clarity purpose (added more clarity in title, and programming notes) as well as some Tables and Listings are clubbed for better presentation, and hence due to that number of the tables, listings and figures are changed.

GlaxoSmithKline Research & Development Limited 205820

Final 1.0

16/Apr/2018

### Statistical Analysis Plan Addendum

#### 2.2 Study objective and secondary end point

In the final SAP Section **2.2** in the secondary objective section of part 2 is stated that secondary endpoint is predose concentration on days 2 to 11. However, for the final analyses secondary endpoint is considered as pre-dose concentration on day 3 to 11.

#### 2.3 Study Design

In the final SAP Section 2.3 in treatment assignment section it is stated that Part 2 treatment section states as below:

"Part 2 treatments:

Treatment D = GSK2838232 500 mg (as 5 x 100 mg) tablet formulation, fed, normal fat (i.e., approximately 30%) meal (reference).

Treatment E = Placebo

However this should be like this:

"Part 2 treatments:

Treatment  $R = GSK2838232\ 500\ mg$  (as 5 x 100 mg) tablet formulation, fed, normal fat (i.e., approximately 30%) meal.

Treatment P = Placebo

#### 2.4 Statistical Hypothesis/Statistical Analysis

For Part 2 study state assessment in the RAP section 2.4 it is stated as below:

Mean plasma GSK2838232 pre-dose values between Days 2 through 11 and  $C\tau$  of Day 11 will be plotted against time.

However it should be as below:

Mean plasma GSK2838232 pre-dose values between Days 3 through 11 and  $C\tau$  of Day 11 will be plotted against time.

#### 2.5 Study Treatment and Sub-group Display Descriptors

In the RAP Section 5.1 Part 2 treatment group descriptors are given as below:

GlaxoSmithKline Research & Development Limited 205820

Final 1.0

16/Apr/2018

TP-EP.BS-WW-008-04 Effective date: 29 Jul 15

# Statistical Analysis Plan Addendum

| Treatment Group Descriptions – Part 2 | | | |
|---|---|---|---|
| | RandAll NG Data Displays for Reporting | | |
| Code | Description | Description | Order in TFL |
| Т3 | GSK2838232 500 mg (as 5 x 100 mg) tablet formulation, fed, normal fat (i.e., approximately 30%) meal (reference). | GSK 500 mg/r tablet fed | 2 |
| P | Placebo | Placebo | 1 |

However it should be as follows:

GlaxoSmithKline Research & Development Limited 205820

Final 1.0

16/Apr/2018

### Statistical Analysis Plan Addendum

| Treatment Group Descriptions – Part 2 | | | |
|---|---|---|---|
| | RandAll NG Data Displays for Reporting | | |
| Code | Description | Description | Order in<br>TFL |
| Т3 | GSK2838232 500 mg (as 5 x 100 mg) tablet formulation, fed, normal fat (i.e., approximately 30%) meal (reference). | GSK 500 mg tablet fed | 2 |
| P | Placebo | Placebo | 1 |

#### 2.6 Concomitant Medications

As per RAP Section 6.4 it is stated that "in the summary of concomitant medications, the ingredients will be summarized by the base only, using CMBASECD and CMBASE". However this is not followed.

#### 2.7 Treatment Compliance and Protocol Deviations

In RAP Section 6.5 it is stated below:

"Information of each participant not received the correct treatment during each treatment period, the reason for not receiving the correct treatment, and any other protocol deviations will be summarized by treatment sequence/group and overall of each part, and listed by participant and period (treatment). In addition, a listing will be provided including dose administered along with dosing dates and time for the investigational product. However it should be as below:

Information of each participant not received the correct treatment during each treatment period, the reason for not receiving the correct treatment, and any other important protocol deviations will be summarized by treatment and overall of each part if enough important protocol deviations occur, and listed by participant and period (treatment). In addition, a listing will be provided including dose administered along with dosing dates and time for the investigational product.

#### 2.8 Derived Pharmacokinetic Parameters

In final RAP section 9.1.1.2, details of derived pharmacokinetic parameter are given as follows:

| Parameter | Parameter Description |
|---|---|
| AUC(0-τ) | Area under the plasma drug concentration-time curve from pre-dose to the end of the dosing interval (where $\tau$ = 24 h) (Day 1 and Day 11) |
| AUC(0-∞) | Area under the concentration-time curve extrapolated to infinity will be calculated as: |
| | $AUC = AUC(0-last) + C(last) / lambda_z$ |

GlaxoSmithKline Research & Development Limited 205820

Final 1.0

16/Apr/2018

TP-EP.BS-WW-008-04 Effective date: 29 Jul 15

### Statistical Analysis Plan Addendum

| Parameter | Parameter Description |
|---|---|
| Cmax | Maximum observed concentration, determined directly from the concentration-time data. (Day 1 and Day 11) |
| Tmax | Time of occurrence of Cmax, determined directly from the concentration-time data (Day 1 and Day 11) |
| Tlag | Lag-time (time delay between drug administration and first observed concentration), determined directly from the concentration-time data (Day 1) |
| Tlast | Time of last quantifiable concentration, determined directly from the concentration-time data (Day 11) |
| t½ | Apparent terminal phase half-life, calculated as; t½ = ln2 / lambda_z (Day 11) |
| Ст | Observed concentration at the end of the dosing interval, determined directly from the concentration-time data (where $\tau = 24$ h) (Day 1 and Day 11) |
| Ctrough | Observed pre-dose concentrations on Days 3 to 11, determined directly from the concentration-time data |

NOTES: C24,  $C\tau$  and Ctrough will be extracted from the concentration data by Clinical Statistics group and merged with other calculated PK parameters provided by CPMS.

All the derived parameters described above will be listed. For each of these parameters, except tmax and tlag, the following summary statistics will be calculated for each treatment group: n, arithmetic mean, standard deviation (SD), median, minimum, maximum, geometric mean with associated 90% CI, standard deviation of logarithmically transformed data, and the between-participant CV (%CVb) based on the geometric mean for the loge-transformed PK parameters. For tmax and tlag, N, n, median, maximum, minimum, arithmetic mean and standard deviation will be calculated.

#### However this should be as below:

| Parameter | Parameter Description |
|---|---|
| AUC(0-τ) | Area under the plasma drug concentration-time curve from pre-dose to the end of the dosing interval (where $\tau$ = 24 h) (Day 1 and Day 11) |
| AUC(0-∞) | Area under the concentration-time curve extrapolated to infinity will be calculated as: $AUC = AUC(0-last) + C(last) / lambda_z$ |
| Cmax | Maximum observed concentration, determined directly from the concentration-time data. (Day 1 and Day 11) |
| Tmax | Time of occurrence of Cmax, determined directly from the concentration-time data (Day 1 and Day 11) |
| Tlag | Lag-time (time delay between drug administration and first observed concentration), determined directly from the concentration-time data (Day 1) |
| Tlast | Time of last quantifiable concentration, determined directly from the concentration-time data (Day 11) |
| t½ | Apparent terminal phase half-life, calculated as; $t\frac{1}{2} = \ln 2 / \text{lambda} z \text{ (Day 11)}$ |
| Сτ | Observed concentration at the end of the dosing interval, determined directly from the |

GlaxoSmithKline Research & Development Limited 205820

Final 1.0

16/Apr/2018

TP-EP.BS-WW-008-04 Effective date: 29 Jul 15

### Statistical Analysis Plan Addendum

| Parameter | Parameter Description |
|---|---|
| | concentration-time data (where $\tau = 24 \text{ h}$ ) (Day 1 and Day 11) |

NOTES: C24, and Cτ will be extracted from the concentration data by Clinical Statistics group and merged with other calculated PK parameters provided by CPMS.

All the derived parameters described above will be listed. For each of these parameters, except tmax and tlag, the following summary statistics will be calculated for each treatment group: N, n, arithmetic mean, standard deviation (SD), median, minimum, maximum, geometric mean with associated 95% CI, standard deviation of logarithmically transformed data, and the between-participant CV (%CVb) based on the geometric mean for the loge-transformed PK parameters. For tmax and tlag, N, n, median, maximum, minimum, arithmetic mean and standard deviation will be calculated.

#### 2.9 Statistical Analysis/Method

#### Part 2

| Parameter | Parameter Description |
|---|---|
| Ctrough | Observed pre-dose concentrations on Days 3 to 11, determined directly from the concentration-time data |
| Ro[AUC(0-<br>τ)] | Accumulation ratio based on AUC(0- $\tau$ ), determined by; Day 11 AUC(0- $\tau$ ) / Day 1 AUC(0- $\tau$ ) |
| R(Cmax) | Accumulation ratio based on Cmax, determined by; Day 11 Cmax / Day 1 Cmax |
| R(Cτ) | Accumulation ratio based on Cτ, determined by; Day 11 Cτ / Day 1 Cτ |

#### NOTES:

- Additional parameters may be included as required.
- Cτ, and Ctrough will be extracted from the concentration data by Clinical Statistics group and merged with other calculated PK parameters provided by CPMS.

All the derived parameters described above will be listed. For each of these parameters, except tmax and tlag, the following summary statistics will be calculated for each treatment group: n, arithmetic mean, standard deviation (SD), median, minimum, maximum, geometric mean with associated 90% CI, standard deviation of logarithmically transformed data, and the between-participant CV (%CVb) based on the geometric mean for the loge-transformed PK parameters. For tmax and tlag, N, n,median, maximum, minimum, arithmetic mean and standard deviation will be calculated.

However is should be as follows:

#### Part 2

| Parameter | Parameter Description |
|---|---|
| Ro[AUC(0-τ)] | Accumulation ratio based on AUC(0- $\tau$ ), determined by; Day 11 AUC(0- $\tau$ ) / Day 1 AUC(0- $\tau$ ) |

GlaxoSmithKline Research & Development Limited 205820

Final 1.0

16/Apr/2018

TP-EP.BS-WW-008-04 Effective date: 29 Jul 15

### Statistical Analysis Plan Addendum

| Parameter | Parameter Description |
|---|---|
| R(Cmax) | Accumulation ratio based on Cmax, determined by; Day 11 Cmax / Day 1 Cmax |
| R(Cτ) | Accumulation ratio based on $C\tau$ , determined by; Day 11 $C\tau$ / Day 1 $C\tau$ |

#### NOTES:

- Additional parameters may be included as required.
- Cτ will be extracted from the concentration data by Clinical Statistics group and merged with other calculated PK parameters provided by CPMS.

All the derived parameters described above will be listed. For each of these parameters, except tmax and tlag, the following summary statistics will be calculated for each treatment group: N, n, arithmetic mean, standard deviation (SD), median, minimum, maximum, geometric mean with associated 95% CI, standard deviation of logarithmically transformed data, and the between-participant CV (%CVb) based on the geometric mean for the loge-transformed PK parameters. For tmax and tlag, N, n,median, maximum, minimum, arithmetic mean and standard deviation will be calculated.

As per final RAP Section 9.2.5, statistical methodology section of Part 2 Steady State Assessment, end point or variable is given as GSK2838232 pre-dose values between Days 2 through 11, however it should be GSK2838232 pre-dose values between Days 3 through 11.

#### 3. TABLES/LISTINGS/FIGURES

#### 3.1 Final Tables, Listings and Figures

Final Table, Listings and Figures that are used for the Final SAC deliverables are shown in tables 1 to 7 for Study Population Tables, Safety Tables, Safety Figures, Pharmacokinetic Tables, Pharmacokinetic Figures, ICH Listings and Non-ICH Listings respectively. The last column "Any Change from the RAP" specifies whether there is any change from RAP for respective Table, Listing or Figure.

Overview of changes from the RAP in final Tables, Listings and Figures are given in tables 8 to 14 for Study Population Tables, Safety Figures, Pharmacokinetic Tables, Pharmacokinetic Figures, ICH Listings and Non-ICH Listings respectively.

Tables 8 to 14 contain only the Tables, Listings and Figures which has any changes from the RAP. Column apart from "Changes from RAP" contains the details from the final RAP.

GlaxoSmithKline Research & Development Limited 205820

Final 1.0

16/Apr/2018

# Statistical Analysis Plan Addendum

Table 1 Study Population Tables

| No | Population | IDSL<br>Shell/TST<br>ID<br>/Example<br>shell | Title | Programming Note | Any<br>Changes<br>in<br>existing<br>RAP |
|---|---|---|---|---|---|
| 1.1 | Safety | ES8A | Summary of Participant<br>Status and Reason for Study<br>Withdrawal – Part 1 | ICH E3, FDAAA,<br>EudraCT<br>Summarize by treatment<br>/sequence and overall of<br>each part | No |
| 1.2 | Safety | ES8 | Summary of Participant<br>Status and Reason for Study<br>Withdrawal – Part 2 | ICH E3, FDAAA,<br>EudraCT<br>Summarize by treatment<br>/sequence and overall of<br>each part | No |
| 1.3 | Safety | SD1 | Summary of Treatment<br>Status and Reasons for<br>Discontinuation of Study<br>Treatment – Part 1 | ICH E3 Summarize by treatment /sequence and overall of each part | No |
| 1.4 | Safety | SD1 | Summary of Treatment<br>Status and Reasons for<br>Discontinuation of Study<br>Treatment – Part 2 | ICH E3 Summarize by treatment /sequence and overall of each part | No |
| 1.5 | Safety | ES4 | Summary of Participant Disposition at Each Study Epoch – Part 1 | ICH E3 | No |
| 1.6 | Safety | ES4 | Summary of Participant Disposition at Each Study Epoch – Part 2 | ICH E3 | No |
| 1.7 | Screened | ES6 | Summary of Screening<br>Status and Reasons for<br>Screen Failure – Part 1 | Journal Requirements | No |
| 1.8 | Screened | ES6 | Summary of Screening<br>Status and Reasons for<br>Screen Failure – Part 2 | Journal Requirements | No |
| 1.9 | Safety | DV1 | Summary of Important<br>Protocol Deviations – Part 1 | ICH E3. If important protocol deviation events are less than 15, please produce the summary with wording"not enough | Yes |

GlaxoSmithKline Research & Development Limited 205820

Final 1.0

16/Apr/2018

TP-EP.BS-WW-008-04 Effective date: 29 Jul 15

# Statistical Analysis Plan Addendum

| | | | | important protocol<br>deviation to warren a<br>summary". | |
|---|---|---|---|---|---|
| 1.10 | Safety | DV1 | Summary of Important<br>Protocol Deviations – Part 2 | ICH E3. If important protocol deviation events are less than 15, please produce the summary with wording not enough important protocol deviation to warren a summary". | Yes |
| 1.11 | Screened | SP1 | Summary of Study<br>Populations – Part 1 | By treatment and combined overall | No |
| 1.12 | Screened | SP1 | Summary of Study<br>Populations – Part 2 | By treatment and combined overall | No |
| 1.13 | Safety | DM3 | Summary of Demographic<br>Characteristics – Part 1 | ICH E3, FDAAA,<br>EudraCT | No |
| 1.14 | Safety | DM1 | Summary of Demographic<br>Characteristics – Part 2 | ICH E3, FDAAA,<br>EudraCT | No |
| 1.15 | Safety | DM11 | Summary of Age Ranges –<br>Part 1 | EudraCT | No |
| 1.16 | Safety | DM11 | Summary of Age Ranges –<br>Part 2 | EudraCT | No |
| 1.17 | Safety | DM5 | Summary of Race and<br>Racial Combinations – Part<br>1 | ICH E3, FDA, FDAAA,<br>EudraCT | No |
| 1.18 | Safety | DM5 | Summary of Race and<br>Racial Combinations – Part<br>2 | ICH E3, FDA, FDAAA,<br>EudraCT | No |
| 1.19 | Safety | MH4 | Summary of Medical<br>Conditions – Part 1 | ICH E3 | No |
| 1.20 | Safety | MH4 | Summary of Medical<br>Conditions – Part 2 | ICH E3 | No |
| 1.21 | Safety | CM8 | Summary of Concomitant<br>Medications – Part 1 | ICH E3 | No |
| 1.22 | Safety | CM8 | Summary of Concomitant<br>Medications – Part 2 | ICH E3 | No |
| 1.23 | Safety | EX1 | Summary of Exposure to<br>Study Treatment – Part 1 | ICH E3 | No |
| 1.24 | Safety | EX1 | Summary of Exposure to<br>Study Treatment – Part 2 | ICH E3 | No |

GlaxoSmithKline Research & Development Limited 205820

Final 1.0

16/Apr/2018

TP-EP.BS-WW-008-04 Effective date: 29 Jul 15

# Statistical Analysis Plan Addendum

Table 2Safety Tables

| No | Population | IDSL<br>Shell/TST<br>ID<br>/Example<br>shell | Title | Programming Note | Any<br>Changes in<br>existing RAP |
|---|---|---|---|---|---|
| 3.1 | Safety | AE5A | Summary of All Adverse<br>Events by Maximum<br>Intensity by System Organ<br>Class and Preferred Term –<br>Part 1 | ICH E3<br>Use AE5A/B (with a<br>Total column across all<br>grades/severities.) | No |
| 3.2 | Safety | AE5A | Summary of All Adverse<br>Events by Maximum<br>Intensity by System Organ<br>Class and Preferred Term –<br>Part 2 | ICH E3 Use AE5A/B (with a Total column across all grades/severities.) | No |
| 3.3 | Safety | AE3 | Summary of Common (>=5%) Adverse Events by Overall Frequency – Part 1 | ICH E3 | No |
| 3.4 | Safety | AE3 | Summary of Common (>=5%) Adverse Events by Overall Frequency – Part 2 | ICH E3 | No |
| 3.5 | Safety | AE5A | Summary of All Drug-<br>Related Adverse Events by<br>System Organ Class and<br>Preferred Term and<br>Maximum Intensity – Part 1 | ICH E3 | No |
| 3.6 | Safety | AE5A | Summary of All Drug-<br>Related Adverse Events by<br>System Organ Class and<br>Preferred Term and<br>Maximum Intensity – Part 2 | ICH E3 | No |
| 3.7 | Safety | AE15 | Summary of Common<br>(>=5%) Non-serious<br>Adverse Events by System<br>Organ Class and Preferred<br>Term (Number of<br>Participant and<br>Occurrences) – Part 1 | FDAAA, EudraCT | No |
| 3.8 | Safety | AE15 | Summary of Common<br>(>=5%) Non-serious<br>Adverse Events by System<br>Organ Class and Preferred<br>Term (Number of<br>Participant and | FDAAA, EudraCT | No |

GlaxoSmithKline Research & Development Limited 205820

Final 1.0

16/Apr/2018

TP-EP.BS-WW-008-04 Effective date: 29 Jul 15

# Statistical Analysis Plan Addendum

| | | | Occurrences) – Part 2 | | |
|---|---|---|---|---|---|
| 3.9 | Safety | AE3 | Summary of Common<br>(>=5%) Grade 2-4 Adverse<br>Events by Overall<br>Frequency – Part 1 | ICH E3 | No |
| 3.10 | Safety | AE3 | Summary of Common<br>(>=5%) Grade 2-4 Adverse<br>Events by Overall<br>Frequency – Part 2 | ICH E3 | No |
| 3.11 | Safety | AE3 | Summary of Common (>=5%) Drug-Related Grade 2-4 Adverse Events by Overall Frequency – Part 1 | ICH E3 | No |
| 3.12 | Safety | AE3 | Summary of Common (>=5%) Drug-Related Grade 2-4 Adverse Events by Overall Frequency – Part 2 | ICH E3 | No |
| 3.13 | Safety | AE16 | Summary of Serious<br>Adverse Events by System<br>Organ Class and Preferred<br>Term (Number of<br>Participants and<br>Occurrences) – Part 1 | FDAAA, EudraCT | No |
| 3.14 | Safety | AE16 | Summary of Serious<br>Adverse Events by System<br>Organ Class and Preferred<br>Term (Number of<br>Participants and<br>Occurrences) – Part 2 | FDAAA, EudraCT | No |
| 3.15 | Safety | AE1 | Summary of Adverse Events Leading to Permanent Discontinuation of Study Treatment or Withdrawal from Study by System Organ Class and Preferred Term /by Overall Frequency – Part 1 | IDSL | No |
| 3.16 | Safety | AE1 | Summary of Adverse Events Leading to Permanent Discontinuation of Study Treatment or Withdrawal from Study by System Organ Class and Preferred Term /by Overall Frequency – Part 2 | IDSL | No |
| 3.17 | Safety | LB17 | Summary of Worst Case<br>Chemistry Results to<br>Potential Clinical | ICH E3 | No |

GlaxoSmithKline Research & Development Limited 205820

Final 1.0

16/Apr/2018

TP-EP.BS-WW-008-04 Effective date: 29 Jul 15

# Statistical Analysis Plan Addendum

| | | | Importance (PCI) Criteria<br>Post-Baseline Relative to<br>Baseline – Part 1 | | |
|---|---|---|---|---|---|
| 3.18 | Safety | LB17 | Summary of Worst Case<br>Chemistry Results to<br>Potential Clinical<br>Importance (PCI) Criteria<br>Post-Baseline Relative to<br>Baseline – Part 2 | ICH E3 | No |
| 3.19 | Safety | LB1 | Summary of Chemistry<br>Changes from Baseline –<br>Part 1 | ICH E3<br>Includes Baseline<br>values. | No |
| 3.20 | Safety | LB1 | Summary of Chemistry<br>Changes from Baseline –<br>Part 2 | ICH E3<br>Includes Baseline<br>values. | No |
| 3.21 | Safety | LB17 | Summary of Worst Case Hematology Results to Potential Clinical Importance (PCI) Criteria Post-Baseline Relative to Baseline – Part 1 | ICH E3 | No |
| 3.22 | Safety | LB17 | Summary of Worst Case Hematology Results to Potential Clinical Importance (PCI) Criteria Post-Baseline Relative to Baseline – Part 2 | ICH E3 | No |
| 3.23 | Safety | LB1 | Summary of Hematology<br>Changes from Baseline –<br>Part 1 | ICH E3<br>Includes Baseline<br>values. | No |
| 3.24 | Safety | LB1 | Summary of Hematology<br>Changes from Baseline –<br>Part 2 | ICH E3<br>Includes Baseline<br>values. | No |
| 3.25 | Safety | LB15 | Summary of Worst Case<br>Urine Data Results Relative<br>to Normal Range Criteria<br>Post-Baseline Relative to<br>Baseline – Part 1 | ICH E3 | No |
| 3.26 | Safety | LB15 | Summary of Worst Case<br>Urine Data Results Relative<br>to Normal Range Criteria<br>Post-Baseline Relative to<br>Baseline – Part 2 | ICH E3 | No |
| 3.27 | Safety | LB1 | Summary of Urine Changes<br>from Baseline – Part 1 | ICH E3<br>Includes Baseline<br>values. | No |

GlaxoSmithKline Research & Development Limited 205820

Final 1.0

16/Apr/2018

TP-EP.BS-WW-008-04 Effective date: 29 Jul 15

# Statistical Analysis Plan Addendum

| 1 | 1 | | 1 | 1 | 1 |
|---|---|---|---|---|---|
| 3.28 | Safety | LB1 | Summary of Urine Changes<br>from Baseline– Part 2 | ICH E3<br>Includes Baseline<br>values. | No |
| 3.29 | Safety | LB1 | Summary of Grade 1 or<br>Higher Lab Abnormalities—<br>Part 1 | Summary of Treatment<br>Emergent Lab toxicity<br>only. | No |
| 3.30 | Safety | LB1 | Summary of Grade 1 or<br>Higher Lab Abnormalities –<br>Part 2 | Summary of Treatment<br>Emergent Lab toxicity<br>only. | No |
| 3.31 | Safety | LIVER1 | Summary of Liver<br>Monitoring/Stopping Event<br>Reporting – Part 1 | IDSL | No |
| 3.32 | Safety | LIVER1 | Summary of Liver<br>Monitoring/Stopping Event<br>Reporting – Part 1 | IDSL | No |
| 3.33 | Safety | LIVER10 | Summary of Subjects Meeting Emergent Hepatobiliary Laboratory Abnormalities Event Reporting – Part 1 | IDSL | No |
| 3.34 | Safety | LIVER10 | Summary of Subjects Meeting Emergent Hepatobiliary Laboratory Abnormalities Event Reporting – Part 2 | IDSL | No |
| 3.35 | Safety | EG1 | Summary of ECG Findings —Part 1 | IDSL Use ECG findings categories (and change from baseline categories, if applicable). | No |
| 3.36 | Safety | EG1 | Summary of ECG Findings —Part 2 | IDSL Use ECG findings categories (and change from baseline categories, if applicable). | No |
| 3.37 | Safety | EG2 | Summary of Change from<br>Baseline in ECG Values—<br>Part 1 | IDSL<br>Includes Baseline<br>values. | No |
| 3.38 | Safety | EG2 | Summary of Change from<br>Baseline in ECG Values—<br>Part 2 | IDSL<br>Includes Baseline<br>values. | No |
| 3.39 | Safety | EG1 | Summary of Category of QTc Data–Part 1 | IDSL | No |
| 3.40 | Safety | EG1 | Summary of Category of | IDSL | No |

GlaxoSmithKline Research & Development Limited 205820

Final 1.0

16/Apr/2018

TP-EP.BS-WW-008-04 Effective date: 29 Jul 15

# Statistical Analysis Plan Addendum

| | | | QTc Data–Part 2 | | |
|---|---|---|---|---|---|
| 3.41 | Safety | EG1 | Summary of Category of<br>QTc Change from Baseline—<br>Part 1 | IDSL<br>Includes Baseline<br>values. | No |
| 3.42 | Safety | EG1 | Summary of Category of<br>QTc Change from Baseline<br>–Part 2 | IDSL<br>Includes Baseline<br>values. | No |
| 3.43 | Safety | VS1 | Summary of Vital Signs –<br>Part 1 | ICH E3 | No |
| 3.44 | Safety | VS1 | Summary of Vital Signs –<br>Part 2 | ICH E3 | No |
| 3.45 | Safety | VS1 | Summary of Change from<br>Baseline in Vital Signs –<br>Part 1 | ICH E3<br>Includes Baseline<br>values. | No |
| 3.46 | Safety | VS1 | Summary of Change from<br>Baseline in Vital Signs –<br>Part 2 | ICH E3 Includes Baseline values. | No |

GlaxoSmithKline Research & Development Limited 205820

Final 1.0

16/Apr/2018

# Statistical Analysis Plan Addendum

### Table 3Safety Figures

| No | Population | IDSL<br>Shell/TST<br>ID<br>/Example<br>shell | Title | Programming Note | Any<br>Changes<br>in<br>existing<br>RAP |
|---|---|---|---|---|---|
| 3.1 | Safety | As EG9 | Plot of Selected Clinical<br>Lab Tests Mean (95% CI)<br>Change from Baseline by<br>Treatment and Time – Part<br>1 | Only include scheduled visits<br>and for selected lab test<br>(BNP, Tnp1, ALT, AST,<br>Bili)<br>Plots will be presented with<br>treatment groups overlaid | Yes |
| 3.2 | Safety | As EG9 | Plot of Selected Clinical<br>Lab Tests Mean (95% CI)<br>Change from Baseline by<br>Treatment and Time – Part<br>2 | Only include scheduled visits<br>and for selected lab test<br>(BNP, Tnp1, ALT, AST,<br>Bili)<br>Plots will be presented with<br>treatment groups overlaid | Yes |
| 3.3 | Safety | EG9 | Plot of Mean (95% CI) Change from Baseline QTcB and QTcF Data by Treatment and Time – Part 1 | Plots will be presented with treatment groups overlaid | Yes |
| 3.4 | Safety | EG9 | Plot of Mean (95% CI)<br>Change from Baseline<br>QTcB and QTcF Data by<br>Treatment and Time – Part<br>2 | Plots will be presented with treatment groups overlaid | Yes |
| 3.5 | Safety | As EG8 | Box Plot of Change from<br>Baseline for Vital Signs by<br>Treatment and Time – Part<br>1 | Plots will be presented with treatment groups overlaid | No |
| 3.6 | Safety | As EG8 | Box Plot of Change from<br>Baseline for Vital Signs by<br>Treatment and Time – Part<br>2 | Plots will be presented with treatment groups overlaid | No |

GlaxoSmithKline Research & Development Limited 205820

Final 1.0

16/Apr/2018

# Statistical Analysis Plan Addendum

#### Table 4 Pharmacokinetic Tables

| No | Population | IDSL<br>Shell/TST ID<br>/Example<br>shell | Title | Programming Note | Any<br>Changes in<br>existing<br>RAP |
|---|---|---|---|---|---|
| 5.1 | PK | PK14 | Listing of Derived Plasma<br>GSK2838232 PK<br>Parameters – Part 1 | Sort by participant and treatment | Yes |
| 5.2 | PK | PK13 | Listing of Derived Plasma<br>GSK2838232 PK<br>Parameters – Part 2 | Sort by participant and treatment | No |
| 5.3 | PK | PK01 | Summary Statistics of<br>Plasma GSK2838232 PK<br>Concentration-Time Data,<br>Bioavailability | | No |
| 5.4 | PK | PK04 | Summary Statistics of<br>Derived Plasma<br>GSK2838232 PK<br>Parameters by Treatment,<br>Bioavailability | | No |
| 5.5 | PK | PK05 | Summary Statistics of<br>Log <sub>e</sub> -transformed Derived<br>Plasma GSK2838232 PK<br>Parameters, Bioavailability | | No |
| 5.6 | PK | Non-Standard1 | Summary of Result of<br>Plasma GSK2838232 PK<br>Parameter Treatment<br>Comparisons for Relative<br>Bioavailability | PK Parameter:<br>AUC(0-inf), and<br>Cmax<br>Ratio: Tablet/Capsule | No |
| 5.7 | PK | PK15 | Listing of Individual Derived Plasma GSK2838232 PK Parameters Treatment Ratios | | No |
| 5.8 | PK | PK01 | Summary Statistics of<br>Plasma GSK2838232 PK<br>Concentration-Time Data,<br>Food Effect | | No |
| 5.9 | PK | PK04 | Summary Statistics of<br>Derived Plasma<br>GSK2838232 PK<br>Parameters by Treatment,<br>Food Effect | | No |
| 5.10 | PK | PK05 | Summary Statistics of<br>Log <sub>e</sub> -transformed Derived<br>Plasma GSK2838232 PK | | No |

GlaxoSmithKline Research & Development Limited 205820

Final 1.0

16/Apr/2018

TP-EP.BS-WW-008-04 Effective date: 29 Jul 15

# Statistical Analysis Plan Addendum

| | | | Parameters, Food Effect | | |
|---|---|---|---|---|---|
| 5.11 | PK | Non-Standard2 | Summary of Result of<br>Plasma GSK2838232 PK<br>Parameter Treatment<br>Comparisons for Food<br>Effect | | No |
| 5.12 | PK | Non-Standard<br>6 | Summary of Result of<br>Plasma GSK2838232 PK<br>Parameter Treatment<br>Comparisons for Food<br>Effect (Non-parametric) | PK Parameter Tmax | Yes |
| 5.13 | PK | PK15 | Listing of Individual Derived Plasma GSK2838232 PK Parameters Treatment Ratios | PK Parameter:<br>AUC(0-inf), Cmax,<br>and tmax<br>Ratio: Fed/Fasted | No |
| 5.14 | PK | PK01 | Summary Statistics of<br>Plasma GSK2838232 PK<br>Concentration-Time Data –<br>Part 2 | Day 1 & Day 11 | No |
| 5.15 | PK | PK04 | Summary Statistics of Derived Plasma GSK2838232 PK Parameters by Treatment and by Day – Part 2 | Day 1 & Day 11 | No |
| 5.16 | PK | PK05 | Summary of Log <sub>e</sub> -<br>transformed Derived<br>Plasma GSK2838232 PK<br>Parameters by Treatment<br>and by Day – Part 2 | Day 1 & Day 11 | No |
| 5.17 | PK | Non-Standard3 | Summary of Results of<br>GSK2838232 PK<br>Parameter Treatment<br>Comparisons -<br>Accumulation<br>Assessments- Part 2 | One for each treatment | No |
| 5.18 | PK | Non-Standard4 | Summary Results of<br>Steady State GSK2838232<br>Concentrations<br>Assessments- Part 2 | One for each treatment | No |

GlaxoSmithKline Research & Development Limited 205820

Final 1.0

16/Apr/2018

# Statistical Analysis Plan Addendum

Table 5 Pharmacokinetic Figures

| No | Population | IDSL<br>Shell/TST ID<br>/Example<br>shell | Title | Programming Note | Any<br>Changes<br>in<br>existing<br>RAP |
|---|---|---|---|---|---|
| 5.1 | PK | PK16B | Individual Plasma GSK2838232 PK Concentration-Time Plots for Relative Bioavailability | Linear and Semi-Log<br>Scale By participant, overlay<br>all treatments for each<br>participant Include LOQ line in plot | Yes |
| 5.2 | PK | PK17 | Mean Plasma GSK2838232<br>PK Concentration for<br>Relative Bioavailability | Linear and Semi-Log<br>Scale<br>Overlay all treatments<br>Include LOQ line in plot | Yes |
| 5.3 | PK | PK18 | Median Plasma GSK2838232 PK Concentration for Relative Bioavailability | Linear and Semi-Log<br>Scale<br>Overlay all treatments<br>Include LOQ line in plot | Yes |
| 5.4 | PK | PK28 | Geometric Mean Treatment<br>Ratio and 90% Confidence<br>Interval of GSK2838232 PK<br>Parameter for the Relative<br>Bioavailability | | No |
| 5.5 | PK | PK25 | Comparative Plot of Individual Plasma GSK2838232 PK Parameters for Relative Bioavailability by treatment | | No |
| 5.6 | PK | PK16A | Individual Plasma<br>GSK2838232 PK<br>Concentration-Time Plots<br>for Food Effect | Linear and Semi-Log<br>Scale<br>By participant, overlay<br>all treatments for each<br>participant<br>Include LOQ line in plot | Yes |
| 5.7 | PK | PK17 | Mean Plasma GSK2838232<br>PK Concentration for Food<br>Effect | Linear and Semi-Log<br>Scale<br>Overlay all treatments<br>Include LLQ line in plot | Yes |
| 5.8 | PK | PK18 | Median Plasma<br>GSK2838232 PK<br>Concentration for Food | Linear and Semi-Log<br>Scale<br>Overlay all treatments | Yes |

GlaxoSmithKline Research & Development Limited 205820

Final 1.0

16/Apr/2018

TP-EP.BS-WW-008-04 Effective date: 29 Jul 15

# Statistical Analysis Plan Addendum

| | | | Effect | Include LOQ line on plot | |
|---|---|---|---|---|---|
| 5.9 | PK | PK28 | Geometric Mean Treatment<br>Ratio and 90% Confidence<br>Interval of GSK2838232 PK<br>Parameter for Food Effect | | No |
| 5.10 | PK | PK25 | Comparative Plot of<br>Individual Plasma<br>GSK2838232 PK<br>Parameters for Food Effect<br>by treatment | | No |
| 5.11 | PK | PK16a | Individual Plasma<br>GSK2838232 PK<br>Concentration-Time Plots by<br>Day – Part 2 | Linear and Semi-Log<br>Scale By participant, overlay<br>days for each participant<br>Include LLQ line on plot | Yes |
| 5.12 | PK | PK17 | Mean Plasma GSK2838232<br>PK Concentration by Day –<br>Part 2 | Linear and Semi-Log<br>Scale<br>Include LLQ line on plot<br>Plot Day 1 and Day 11<br>on Separate page | Yes |
| 5.13 | PK | PK18 | Median Plasma<br>GSK2838232 PK<br>Concentration by Day – Part<br>2 | Linear and Semi-Log<br>Scale<br>Include LLQ line on plot<br>Plot Day 1 and Day 11<br>on Separate page | Yes |
| 5.14 | PK | PK16a | Individual Plasma GSK2838232 Predose Concentration-Time Plots for Steady State Assessment – Part 2 | Linear and Semi-Log Scale Overlay all individual profile with all days profiles Day on x-axis, predose concentration on y-axis, join day to day for each subject. | Yes |
| 5.15 | PK | PK17 | Mean Plasma GSK2838232<br>Concentration-Time Plots<br>for Steady State Assessment<br>– Part 2 | Linear and Semi-Log Scale Days on same plot with x-axis as Days, mean concentration plotted across and joined | Yes |
| 5.16 | PK | PK18 | Median Plasma<br>GSK2838232<br>Concentration-Time Plots<br>for Steady State Assessment<br>– Part 2 | Linear and Semi-Log Scale Days on same plot with x-axis as Days, median concentration plotted across and joined | Yes |

GlaxoSmithKline Research & Development Limited 205820

Final 1.0

16/Apr/2018

TP-EP.BS-WW-008-04 Effective date: 29 Jul 15

# Statistical Analysis Plan Addendum

| 5.17 | PK | PK16a | Individual and Box Plot of | Include all the PK | Yes |
|---|---|---|---|---|---|
| | | | Plasma GSK2838232 PK | parameters. | |
| | | | Parameters by Day – Part 2 | | |
| 5.18 | PK | PK25 | Comparative Plot of Plasma<br>GSK2838232 PK<br>Parameters for<br>Accumulation | Linear and Log Scale | Yes |

GlaxoSmithKline Research & Development Limited 205820

Final 1.0

16/Apr/2018
# Statistical Analysis Plan Addendum

## Table 6 ICH Listings

| No | Population | IDSL<br>Shell/TST<br>ID<br>/Example<br>shell | Title | Programming Note | Any<br>Changes<br>in<br>existing<br>RAP |
|---|---|---|---|---|---|
| 1 | Screened | ES7 | Listing of Reasons for Screen<br>Failure – Part 1 | | No |
| 2 | Screened | ES7 | Listing of Reasons for Screen<br>Failure – Part 2 | | No |
| 3 | Safety | ES3 | Listing of Reasons for Study<br>Withdrawal – Part 1 | | No |
| 4 | Safety | ES2 | Listing of Reasons for Study<br>Withdrawal – Part 2 | | No |
| 5 | Safety | SD3 | Listing of Reasons for Study<br>Treatment Discontinuation –<br>Part 1 | | No |
| 6 | Safety | SD2 | Listing of Reasons for Study<br>Treatment Discontinuation –<br>Part 2 | | No |
| 7 | Safety | BL1 | Listing of Participants for<br>Whom the Treatment Blind was<br>Broken – Part 2 | | No |
| 8 | Safety | CP_RA1x | Listing of Planned and Actual<br>Treatments – Part 1 | | No |
| 9 | Safety | CP_RA1p | Listing of Planned and Actual<br>Treatments – Part 2 | | No |
| 10 | Safety | DV2A | Listing of Important Protocol<br>Deviations – Part 1 | ICH E3<br>Listing also includes<br>analysis population<br>exclusions. | No |
| 11 | Safety | DV2 | Listing of Important Protocol<br>Deviations – Part 2 | ICH E3 Listing also includes analysis population exclusions. | No |
| 12 | Safety | IE4 | Listing of Participants with Inclusion/Exclusion Criteria Deviations – Part 1 | ICH E3 | No |
| 13 | Safety | IE3 | Listing of Participants with<br>Inclusion/Exclusion Criteria<br>Deviations – Part 2 | ICH E3 | No |
| 14 | Safety | SP3A | Listing of Participants Excluded from Any Population – Part 1 | ICH E3 | No |

GlaxoSmithKline Research & Development Limited 205820

Final 1.0

16/Apr/2018

TP-EP.BS-WW-008-04 Effective date: 29 Jul 15

# Statistical Analysis Plan Addendum

| 15 | Safety | SP3 | Listing of Participants Excluded from Any Population – Part 2 | ICH E3 | No |
|---|---|---|---|---|---|
| 16 | Safety | DM4 | Listing of Demographic<br>Characteristics – Part 1 | ICH E3 | No |
| 17 | Safety | DM2 | Listing of Demographic<br>Characteristics – Part 2 | ICH E3 | No |
| 18 | Safety | DM10 | Listing of Race – Part 1 | ICH E3 | No |
| 19 | Safety | DM9 | Listing of Race – Part 2 | ICH E3 | No |
| 20 | Safety | CP_CM4 | Listing of Concomitant<br>Medications – Part 1 | IDSL | No |
| 21 | Safety | CP_CM3 | Listing of Concomitant<br>Medications – Part 2 | IDSL | No |
| 22 | Safety | EX4 | Listing of Exposure Data – Part 1 | ICH E3 | No |
| 23 | Safety | EX3 | Listing of Exposure Data – Part 2 | ICH E3 | No |
| 24 | Safety | CP_AE9 | Listing of All Adverse Events – Part 1 | ICH E3 | No |
| 25 | Safety | CP_AE8 | Listing of All Adverse Events – Part 2 | ICH E3 | No |
| 26 | Safety | AE7 | Listing of Participant Numbers<br>for Individual Adverse Events –<br>Part 1 | ICH E3 | No |
| 27 | Safety | AE7 | Listing of Participant Numbers<br>for Individual Adverse Events –<br>Part 2 | ICH E3 | No |
| 28 | Safety | AE2 | Listing of Relationship Between Adverse Event System Organ Classes, Preferred Terms, and Verbatim Text – Part 1 | IDSL | No |
| 29 | Safety | AE2 | Listing of Relationship Between Adverse Event System Organ Classes, Preferred Terms, and Verbatim Text – Part 2 | IDSL | No |
| 30 | Safety | CP_AE9a | Listing of Fatal Serious<br>Adverse Events – Part 1 | ICH E3 | No |
| 31 | Safety | CP_AE8a | Listing of Fatal Serious<br>Adverse Events – Part 2 | ICH E3 | No |
| 32 | Safety | CP_AE9a | Listing of Non-Fatal Serious<br>Adverse Events – Part 1 | ICH E3 | No |
| 33 | Safety | CP_AE8a | Listing of Non-Fatal Serious | ICH E3 | No |
| | | | - | | |

GlaxoSmithKline Research & Development Limited 205820

Final 1.0

16/Apr/2018

TP-EP.BS-WW-008-04 Effective date: 29 Jul 15

# Statistical Analysis Plan Addendum

| | | | Adverse Events – Part 2 | | |
|---|---|---|---|---|---|
| 34 | Safety | AE14 | Listing of Reasons for<br>Considering as a Serious<br>Adverse Event | ICH E3 | No |
| 35 | Safety | CP_AE9a | Listing of Adverse Events Leading to Withdrawal from Study / Permanent Discontinuation of Study Treatment – Part 1 | ICH E3 | No |
| 36 | Safety | CP_AE8a | Listing of Adverse Events<br>Leading to Withdrawal from<br>Study / Permanent<br>Discontinuation of Study<br>Treatment – Part 2 | ICH E3 | No |
| 37 | Safety | CP_AE9a | Listing of Grade 3 or 4 Adverse<br>Events – Part 1 | Division of AIDS<br>Table For Grading | No |
| 38 | Safety | CP_AE8a | Listing of Grade 3 or 4 Adverse<br>Events – Part 2 | Division of AIDS<br>Table For Grading | No |
| 39 | Safety | MH2 | Listing of Medical Conditions<br>for Participants with Liver<br>Stopping Events – Part 1 | IDSL | No |
| 40 | Safety | MH2 | Listing of Medical Conditions<br>for Participants with Liver<br>Stopping Events – Part 2 | IDSL | No |
| 41 | Safety | SU2 | Listing of Substance Use for<br>Participants with Liver<br>Stopping Events – Part 1 | IDSL | No |
| 42 | Safety | SU2 | Listing of Substance Use for<br>Participants with Liver<br>Stopping Events – Part 2 | IDSL | No |
| 43 | Safety | LB13 | Listing of Reference Ranges for<br>Clinical Laboratory Tests | | No |
| 44 | Safety | LB6 | Listing of Hematology Data–<br>Part 1 | If any laboratory test<br>results are outside of<br>the reference range,<br>they will be flagged<br>with high/low and/or<br>toxicity grade in the<br>listing | No |
| 45 | Safety | LB5 | Listing of Hematology Data–<br>Part 2 | If any laboratory test<br>results are outside of<br>the reference range,<br>they will be flagged<br>with high/low and/or<br>toxicity grade in the<br>listing | No |
| 46 | Safety | LB6 | Listing of Clinical Chemistry | If any laboratory test | No |

GlaxoSmithKline Research & Development Limited 205820

Final 1.0

16/Apr/2018

TP-EP.BS-WW-008-04 Effective date: 29 Jul 15

# Statistical Analysis Plan Addendum

| | | | Data– Part 1 | results are outside of<br>the reference range,<br>they will be flagged<br>with high/low and/or<br>toxicity grade in the<br>listing | |
|---|---|---|---|---|---|
| 47 | Safety | LB5 | Listing of Clinical Chemistry<br>Data– Part 2 | If any laboratory test<br>results are outside of<br>the reference range,<br>they will be flagged<br>with high/low and/or<br>toxicity grade in the<br>listing | No |
| 48 | Safety | LB6 | Listing of Urinalysis Data– Part 1 | If any laboratory test<br>results are outside of<br>the reference range,<br>they will be flagged<br>with high/low and/or<br>toxicity grade in the<br>listing | No |
| 49 | Safety | LB5 | Listing of Urinalysis Data– Part 2 | If any laboratory test<br>results are outside of<br>the reference range,<br>they will be flagged<br>with high/low and/or<br>toxicity grade in the<br>listing | No |
| 50 | Safety | LB6 | Listing of All Laboratory Data<br>for Participants with Any Value<br>of Potential Clinical<br>Importance—Part 1 | ICH E3 May be split into separate listings by chemistry, hematology, etc. Display ALL labs for a participant who experienced a value of potential clinical importance. | No |
| 51 | Safety | LB5 | Listing of All Laboratory Data<br>for Participants with Any Value<br>of Potential Clinical<br>Importance– Part 2 | ICH E3 May be split into separate listings by chemistry, hematology, etc. Display ALL labs for a participant who experienced a value of potential clinical importance. | No |
| 52 | Safety | LB6 | Listing of Lab Results<br>Identified as Adverse Events— | Lab results identified as AEs. Only needed | No |

GlaxoSmithKline Research & Development Limited 205820

Final 1.0

16/Apr/2018

TP-EP.BS-WW-008-04 Effective date: 29 Jul 15

# Statistical Analysis Plan Addendum

| | | ı | I | | |
|---|---|---|---|---|---|
| | | | Part 1 | if there are a<br>sufficient number of<br>labs identified as<br>AEs. | |
| 53 | Safety | LB5 | Listing of Lab Results<br>Identified as Adverse Events –<br>Part 2 | Lab results identified<br>as AEs. Only needed<br>if there are a<br>sufficient number of<br>labs identified as<br>AEs. | No |
| 54 | Safety | LB6 | Listing of Grade 2 or Higher<br>Lab Abnormalities – Part 1 | | No |
| 55 | Safety | LB5 | Listing of Grade 2 or Higher<br>Lab Abnormalities – Part 2 | | No |
| 56 | Safety | LB14 | Listing of Laboratory Data with<br>Character Results – Part 1 | ICH E3 | No |
| 57 | Safety | LB14 | Listing of Laboratory Data with<br>Character Results – Part 2 | ICH E3 | No |
| 58 | Safety | UR2B | Listing of Urinalysis Data for<br>Participants with Any Value of<br>Potential Clinical Importance –<br>Part 1 | ICH E3 Display ALL data for a participant who experienced a value of potential clinical importance. | No |
| 59 | Safety | UR2A | Listing of Urinalysis Data for<br>Participants with Any Value of<br>Potential Clinical Importance –<br>Part 2 | ICH E3 Display ALL data for a participant who experienced a value of potential clinical importance. | No |
| 60 | Safety | EG4 | Listing of All ECG Values for<br>Participants with Any Value of<br>Potential Clinical Importance –<br>Part 1 | IDSL | No |
| 61 | Safety | EG3 | Listing of All ECG Values for<br>Participants with Any Value of<br>Potential Clinical Importance –<br>Part 2 | IDSL | No |
| 62 | Safety | EG6 | Listing of All ECG Findings for<br>Participants with an Abnormal<br>ECG Finding – Part 1 | IDSL | No |
| 63 | Safety | EG5 | Listing of All ECG Findings for<br>Participants with an Abnormal<br>ECG Finding – Part 2 | IDSL | No |
| 64 | Safety | HM8 | Listing of Holter Monitoring –<br>Part 1 | IDSL | No |

GlaxoSmithKline Research & Development Limited 205820

Final 1.0

16/Apr/2018

TP-EP.BS-WW-008-04 Effective date: 29 Jul 15

# Statistical Analysis Plan Addendum

| 65 | Safety | HM8 | Listing of Holter Monitoring –<br>Part 2 | IDSL | No |
|---|---|---|---|---|---|
| 66 | Safety | VS5 | Listing of All Vital Signs Data<br>for Participants with Any Value<br>of Potential Clinical Importance<br>– Part 1 | IDSL | No |
| 67 | Safety | VS4 | Listing of All Vital Signs Data<br>for Participants with Any Value<br>of Potential Clinical Importance<br>– Part 2 | IDSL | No |
| 68 | Safety | Non-<br>Standard 5 | Listing of Meal- Part 1 | | Yes |

GlaxoSmithKline Research & Development Limited 205820

Final 1.0

16/Apr/2018

# Statistical Analysis Plan Addendum

## Table 7 Non-ICH Lisitngs

| No | Population | IDSL<br>Shell/TST ID<br>/Example shell | Title | Programming Note | Any<br>Changes in<br>existing<br>RAP |
|---|---|---|---|---|---|
| 69 | PK | PK08 | Listing of Plasma GSK2838232 PK Concentration-Time Data -Part 1 | Sort by participant, treatment, day, and time | Yes |
| 70 | PK | PK07 | Listing of Plasma GSK2838232 PK Concentration-Time Data -Part 2 | Sort by participant, treatment, day, and time | Yes |
| 71 | PK | SAS output of<br>Table 5.6 | SAS Output of Summary Results of GSK2838232 PK Parameter Treatment Comparisons for the Relative Bioavailability – Part 1A | | Yes |
| 72 | PK | SAS output of<br>Table 5.10 | SAS Output of Summary<br>Results of GSK2838232<br>PK Parameter Treatment<br>Comparisons for the Food<br>Effect – Part 1B | | Yes |
| 73 | PK | SAS output of<br>Table 5.12 | SAS Output of Summary Results of GSK2838232 PK Parameter Treatment Comparisons for the Food Effect (Non-parametric) – Part 1B | | Yes |
| 74 | PK | SAS output of<br>Table 5.16 | SAS Output of Summary<br>Results of Steady-State<br>GSK2838232<br>Concentrations Assessment<br>– Part 2 | | Yes |
| 75 | PK | SAS output of<br>Table 5.17 | SAS Output of Summary Results of GSK2838232 PK Parameter Treatment Comparisons – Accumulation Ratio – Part 2 | | Yes |

GlaxoSmithKline Research & Development Limited 205820

Final 1.0

# Statistical Analysis Plan Addendum

## Table 8 Study Population Tables (Changes from RAP)

| No | Populatio<br>n | IDSL<br>Shell/TST<br>ID<br>/Example<br>shell | Title | Programming<br>Note | Changes done from the RAP |
|---|---|---|---|---|---|
| 1.9 | Safety | DV1 | Summary of<br>Protocol<br>Deviations – Part 1 | ICH E3 | 1. Title has been changed from "Summary of Protocol Deviations – Part 1" to "Summary of Important Protocol Deviations – Part 1" 2. Programming note has been appended with following texts: "If important protocol deviation events are less than 15, please produce the summary with wordings" not enough important protocol deviation to warren a summary". |
| 1.10 | Safety | DV1 | Summary of<br>Protocol<br>Deviations – Part 2 | ICH E3 | 1. Title has been changed from "Summary of Protocol Deviations – Part 2" to "Summary of Important Protocol Deviations – Part 2" 2. Programming note has been appended with following texts: "If important protocol deviation events are less than 15, please produce the summary with wordings "not enough important protocol deviation to warren a summary". |

GlaxoSmithKline Research & Development Limited 205820

Final 1.0

# Statistical Analysis Plan Addendum

Table 9 Safety Figures (Changes from RAP)

| No | Population | IDSL<br>Shell/TST ID<br>/Example<br>shell | Title | Programming<br>Note | Changes from RAP |
|---|---|---|---|---|---|
| 3.1 | Safety | As EG9 | Plot of Selected Clinical<br>Lab Tests Mean Change<br>from Baseline by<br>Treatment and Time –<br>Part 1 | Only include<br>scheduled visits<br>and for selected<br>lab test (BNP,<br>Tnp1, ALT,<br>AST, Bili)<br>Plots will be<br>presented with<br>treatment<br>groups overlaid | Title has been changed<br>to "Plot of Selected<br>Clinical Lab Tests<br>Mean (95% CI)<br>Change from Baseline<br>by Treatment and<br>Time – Part 1" |
| 3.2 | Safety | As EG9 | Plot of Selected Clinical<br>Lab Tests Mean Change<br>from Baseline by<br>Treatment and Time –<br>Part 2 | Only include<br>scheduled visits<br>and for selected<br>lab test (BNP,<br>Tnp1, ALT,<br>AST, Bili)<br>Plots will be<br>presented with<br>treatment<br>groups overlaid | Title has been changed<br>to "Plot of Selected<br>Clinical Lab Tests<br>Mean (95% CI)<br>Change from Baseline<br>by Treatment and<br>Time – Part 2" |
| 3.3 | Safety | EG9 | Plot of Mean Change<br>from Baseline QTcB and<br>QTcF Data by Treatment<br>and Time – Part 1 | Plots will be<br>presented with<br>treatment<br>groups overlaid | Title has been changed<br>to "Plot of Mean (95%<br>CI) Change from<br>Baseline QTcB and<br>QTcF Data by<br>Treatment and Time –<br>Part 1" |
| 3.4 | Safety | EG9 | Plot of Mean Change<br>from Baseline QTcB and<br>QTcF Data by Treatment<br>and Time – Part 2 | Plots will be<br>presented with<br>treatment<br>groups overlaid | Title has been changed<br>to "Plot of Mean (95%<br>CI) Change from<br>Baseline QTcB and<br>QTcF Data by<br>Treatment and Time –<br>Part 2" |

GlaxoSmithKline Research & Development Limited 205820

Final 1.0

# Statistical Analysis Plan Addendum

## Table 10 Pharmacokinetic Tables (Changes from RAP)

| No | Population | IDSL<br>Shell/TST ID<br>/Example<br>shell | Title | Programming<br>Note | Changes from RAP |
|---|---|---|---|---|---|
| 5.1 | PK | PK14 | Listing of Derived Plasma<br>GSK2838232 PK<br>Parameters – Part<br>1A | Sort by participant and treatment | This table is clubbed with table 5.2 Title has been changed to "Listing of Derived Plasma GSK2838232 PK Parameters – Part 1" |
| 5.2 | PK | PK14 | Listing of Derived Plasma<br>GSK2838232 PK<br>Parameters – Part<br>1B | Sort by participant and treatment | This table has been removed. |
| 5.3 | PK | PK13 | Listing of Derived Plasma<br>GSK2838232 PK<br>Parameters – Part 2 | Sort by participant and treatment | Table no is changed to 5.2 |
| x.xx | PK | Non-Standard<br>6 | Summary of Result of<br>Plasma GSK2838232 PK<br>Parameter Treatment<br>Comparisons for Food<br>Effect (Non-parametric) | PK Parameter<br>Tmax | Newly added, with<br>Table no 5.12 |
| 5.14 | PK | PK04 | Summary Statistics of<br>Plasma GSK2838232 PK<br>Parameters by Treatment<br>and by Day – Part 2 | Day 1 & Day<br>11 | Title has been changed to "Summary Statistics of Plasma GSK2838232 PK Concentration time data by Treatment and by Day – Part 2 |

GlaxoSmithKline Research & Development Limited 205820

Final 1.0

# Statistical Analysis Plan Addendum

Table 11 Pharmacokinetic Figures (Changes from RAP)

| No | Population | IDSL<br>Shell/TST<br>ID<br>/Example<br>shell | Title | Programming<br>Note | Changes from RAP |
|---|---|---|---|---|---|
| 5.1 | PK | PK16B | Individual Plasma GSK2838232 PK Concentration-Time Plots for Relative Bioavailability | Linear and Semi-<br>Log Scale By participant, overlay all treatments for each participant Include LOQ line in plot | In programming note "Include LOQ line in plot" is added |
| 5.2 | PK | PK17 | Mean Plasma GSK2838232<br>PK Concentration for<br>Relative Bioavailability | Linear and Semi-<br>Log Scale<br>Overlay all<br>treatments<br>Include LOQ<br>line in plot | In programming note "Include LOQ line in plot" is added |
| 5.3 | PK | PK18 | Median Plasma GSK2838232 PK Concentration for Relative Bioavailability | Linear and Semi-<br>Log Scale<br>Overlay all<br>treatments<br>Include LOQ<br>line in plot | In programming note "Include LOQ line in plot" is added |
| 5.6 | PK | PK16A | Individual Plasma GSK2838232 PK Concentration-Time Plots for Food Effect | Linear and Semi-<br>Log Scale By participant, overlay all treatments for each participant Include LOQ line in plot | In programming note "Include LOQ line in plot" is added |
| 5.7 | PK | PK17 | Mean Plasma GSK2838232<br>PK Concentration for Food<br>Effect | Linear and Semi-<br>Log Scale<br>Overlay all<br>treatments<br>Include LLQ line<br>in plot | In programming note "Include LOQ line in plot" is added |
| 5.8 | PK | PK18 | Median Plasma GSK2838232 PK Concentration for Food Effect | Linear and Semi-<br>Log Scale<br>Overlay all<br>treatments<br>Include LOQ | In programming note "Include LOQ line in plot" is added |

GlaxoSmithKline Research & Development Limited 205820

Final 1.0

16/Apr/2018

TP-EP.BS-WW-008-04 Effective date: 29 Jul 15

# Statistical Analysis Plan Addendum

| | | | | line on plot | |
|---|---|---|---|---|---|
| 5.11 | PK | PK16a | Individual Plasma GSK2838232 PK Concentration-Time Plots by Day – Part 2 | Linear and Semi-<br>Log Scale<br>By participant,<br>overlay days for<br>each participant<br>Include LLQ line<br>on plot | In programming note "Include LOQ line in plot" is added |
| 5.12 | PK | PK17 | Mean Plasma GSK2838232<br>PK Concentration by Day –<br>Part 2 | Linear and Semi-<br>Log Scale<br>Include LLQ line<br>on plot<br>Plot Day 1 and<br>Day 11 on<br>Separate page | In programming note Include LLQ line on plot Plot Day 1 and Day 11 on Separate page are added. |
| 5.13 | PK | PK18 | Median Plasma GSK2838232 PK Concentration by Day – Part 2 | Linear and Semi-<br>Log Scale<br>Include LLQ line<br>on plot<br>Plot Day 1 and<br>Day 11 on<br>Separate page | In programming note Include LLQ line on plot Plot Day 1 and Day 11 on Separate page are added. |
| 5.19 | PK | PK16a | Individual Plasma GSK2838232 Predose Concentration-Time Plots for Steady State Assessment – Part 2 | Linear and Semi-<br>Log Scale Overlay all individual profile with all days profiles Day on x-axis, predose concentration on y-axis, join day to day for each subject. | In programming note Day on x-axis, predose concentration on y- axis, and join day to day for each subject is added. Figure no change to 5.14 |
| 5.20 | PK | PK17 | Mean Plasma GSK2838232<br>Concentration-Time Plots<br>for Steady State Assessment<br>– Part 2 | Linear and Semi-<br>Log Scale Days on same plot with x-axis as Days, mean concentration plotted across and joined | In programming note<br>Days on same plot<br>with x-axis as Days,<br>mean concentration<br>plotted across and<br>joined, is added.<br>Figure no change 5.15 |
| 5.21 | PK | PK18 | Median Plasma GSK2838232 Concentration-Time Plots for Steady State Assessment – Part 2 | Linear and Semi-<br>Log Scale Days on same plot with x-axis as Days, median concentration | In programming note Days on same plot with x-axis as Days, median concentration plotted across and joined, is added. |

GlaxoSmithKline Research & Development Limited 205820

Final 1.0

16/Apr/2018

TP-EP.BS-WW-008-04 Effective date: 29 Jul 15

# Statistical Analysis Plan Addendum

| | | | | plotted across<br>and joined | Figure no changed to 5.16 |
|---|---|---|---|---|---|
| 5.22 | PK | PK16a | Individual and Box Plot of<br>Plasma GSK2838232 PK<br>Parameters by Day – Part 2 | Include all the PK parameters. | Figure no change to 5.17 |
| 5.23 | PK | PK25 | Comparative Plot of Plasma<br>GSK2838232 PK<br>Parameters for<br>Accumulation | Linear and Log<br>Scale | Figure no change to 5.18 |

GlaxoSmithKline Research & Development Limited 205820

Final 1.0

16/Apr/2018

# Statistical Analysis Plan Addendum

## Table 12 ICH Listing (Changes from RAP)

| No | Population | IDSL<br>Shell/TST ID<br>/Example<br>shell | Title | Programming<br>Note | Changes from<br>RAP |
|---|---|---|---|---|---|
| XX | Safety | Non-Standard<br>5 | Listing of Meal Data - Part | Part 1 only | Newly Added with listing no 68 |

GlaxoSmithKline Research & Development Limited 205820

Final 1.0

16/Apr/2018

# Statistical Analysis Plan Addendum

## Table 13 Non-ICH Listings (Change from RAP)

| No | Population | IDSL<br>Shell/TST<br>ID<br>/Example<br>shell | Title | Programming<br>Note | Changes from RAP |
|---|---|---|---|---|---|
| 68 | PK | PK08 | Listing of Plasma<br>GSK2838232 PK<br>Concentration-<br>Time Data -Part<br>1A | Sort by participant, treatment, day, and time | This listing has been combined with listing number 69. Title of this listing is changed to "Listing of Plasma GSK2838232 PK Concentration-Time Data —Part 1" This listing number has been changed to 69. |
| 69 | PK | PK08 | Listing of Plasma<br>GSK2838232 PK<br>Concentration-<br>Time Data -Part<br>1B | Sort by participant, treatment, day, and time | This listing has been removed |
| xx | PK | SAS<br>output of<br>Table 5.12 | SAS Output of<br>Summary Results<br>of GSK2838232<br>PK Parameter<br>Treatment<br>Comparisons for<br>the Food Effect<br>(Non-parametric) –<br>Part 1B | | This is newly added |
| 73 | PK | SAS<br>output of<br>Table 5.16 | SAS Output of<br>Summary Results<br>of Steady-State<br>GSK2838232<br>Concentrations<br>Assessment – Part<br>2 | | This listing number is changed to 74 |
| 74 | PK | SAS<br>output of<br>Table 5.17 | SAS Output of Summary Results of GSK2838232 PK Parameter Treatment Comparisons – Accumulation Ratio – Part 2 | | This listing no is changed to 75 |

GlaxoSmithKline Research & Development Limited 205820

Final 1.0

16/Apr/2018

TP-EP.BS-WW-008-04 Effective date: 29 Jul 15

# Statistical Analysis Plan Addendum

#### 4. SHELLS

Example: Non-Standard 5

Protocol: AAA111111
Population: Safety

Page 1 of xx

Listing x
Listing of Meal Data (Safety Population)

| {Inv./}<br>Subj. | {Age(y)/<br>Sex/<br>Race} | Trt. | Visit/Pl.<br>Time | Start<br>Date/Star<br>t Time of<br>Meal | • | Start Date/Star t Time of Dosing | | Totality of the Meal been Ingested ? | Proporti onal of the Meal Consumed ? |
|---|---|---|---|---|---|---|---|---|---|
| PPD | 36/ | A | PART1 | PPD | | | High Fat | No | 76- |
| | M/<br>Mixed Race | | P1D1/PRED<br>OSE | /09:00 | 9/09:10 | /09:30 | Meal | | 100% |

GlaxoSmithKline Research & Development Limited 205820

Final 1.0

16/Apr/2018

TP-EP.BS-WW-008-04 Effective date: 29 Jul 15

# Statistical Analysis Plan Addendum

Example: Non-Standard 6

Protocol: AAA111111 Page 1 of xx

Population: Pharmacokinetic

Table x

Summary of Result of Plasma GSK2838232 PK Parameter Treatment Comparisons for Food Effect (Non-Parametric)

| | | Med | ian | | | |
|---|---|---|---|---|---|---|
| PK Parameter | Comparison<br>Test/Ref. | GSK 200 mg/r<br>tablet fasted<br>(N=xx) | GSK 200 mg/r<br>tablet fed<br>(N=xx) | Diffe<br>rence | 90% Confidence<br>Interval | p-value |
| Tmax(h) | GSK 200 mg/r tablet fed<br>vs GSK 200 mg/r tablet<br>fasted | xx.xx | xx.xx | | (xx.xx,xx.xx) | x.xxxx |

GlaxoSmithKline Research & Development Limited 205820

Final 1.0

16/Apr/2018

TP-EP.BS-WW-008-04 Effective date: 29 Jul 15

## Statistical Analysis Plan Addendum

## 5. REFERENCES

- SAS® Version 9.3 of the SAS System for Personal Computers. Copyright © 2002-2003. SAS Institute Inc. SAS and all other SAS Institute Inc. product or service names are registered trademarks or trademarks of SAS Institute Inc., Cary, NC, USA.
- 2. WinNonlin Professional Software Version 5.2. <a href="http://www.pharsight.com">http://www.pharsight.com</a>

GlaxoSmithKline Research & Development Limited 205820

Final 1.0

16/Apr/2018